CLINICAL TRIAL: NCT00856544
Title: Phase 3, Randomized, Double Blind, Placebo Controlled Study Of The Safety And Efficacy Of 2 Doses Of CP 690,550 In Patients With Active Rheumatoid Arthritis On Background DMARDS
Brief Title: A Study Comparing 2 Doses Of CP-690,550 Vs. Placebo For The Treatment Of Rheumatoid Arthritis In Patients On Other Background Arthritis Medications
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921046
Record Dates: First submitted 2009-03-03; First posted 2009-03-05 (Estimated); Results first posted 2013-01-10 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2012-12

CONDITIONS: Arthritis, Rheumatoid
Keywords: Arthritis; Rheumatoid; Antirheumatic Agents; Clinical Trial
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Active 5 mg (Experimental)
  Interventions: Drug: CP-690,550
- Active 10 mg (Experimental)
  Interventions: Drug: CP-690,550
- Placebo Sequence 1 (Placebo Comparator): Placebo non-responders advance to 5 mg CP-690,550 at Month 3 visit. All patients in this treatment arm advance to 5 mg CP-690,550 at Month 6 visit.
  Interventions: Drug: Placebo
- Placebo Sequence 2 (Placebo Comparator): Placebo non-responders advance to 10 mg CP-690,550 at Month 3 visit. All patients in this treatment arm advance to 10 mg CP-690,550 at Month 6 visit.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CP-690,550 — Film coated tablet, 5 mg PO BID, 1 year
  Arms: Active 5 mg
Drug: CP-690,550 — Film coated tablet, 10 mg PO BID, 1 year
  Arms: Active 10 mg
Drug: Placebo — Film coated tablet, 1 tablet PO BID, 3-6 months
  Arms: Placebo Sequence 1
Drug: Placebo — Film coated tablet, 1 tablet PO BID, 3-6 months
  Arms: Placebo Sequence 2

SUMMARY:
This Phase 3 study is intended to provide evidence that CP-690,550 dosed 5 mg BID and 10 mg BID is safe and effective when used in combination with a variety of traditional disease modifying antirheumatic drugs in adult patients with rheumatoid arthritis. It is intended to confirm the benefits of CP-690,550 in improving signs and symptoms and physical function that were observed in the Phase 2 rheumatoid arthritis studies.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a diagnosis of Rheumatoid Arthritis based on the American College of Rheumatology (ACR) 1987 Revised Criteria.
* The patient has active disease as defined by both >=4 tender or painful joints on motion and >= 4 joints swollen; and either an erythrocyte sedimentation rate (ESR) > 28 mm or a C-reactive protein (CRP) concentration > 7 mg/dL.
* Patient had an inadequate response to at least one disease modifying antirheumatic drug (traditional or biologic) due to lack of efficacy or toxicity.
* Patient must remain on at least one background traditional disease modifying antirheumatic drug.
* No evidence of inadequately treated latent or active infection with Mycobacterium tuberculosis.

Exclusion Criteria:

* Blood dyscrasias including confirmed: Hemoglobin <9 g/dL or Hematocrit <30%; White blood cell count <3.0 x 109/L; Absolute neutrophil count <1.2 x 109/L; Platelet count <100 x 109/L.
* History of any other rheumatic autoimmune disease other than Sjogren's syndrome.
* No malignancy or history of malignancy.
* History of infection requiring hospitalization, parenteral antimicrobial therapy, or as otherwise judged clinically significant by the investigator, within the 6 months prior to the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 795 (Actual)
Dates: Start 2009-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (122):
- United States (44):
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Jonesboro, Arkansas
  - Pfizer Investigational Site, Palo Alto, California
  - Pfizer Investigational Site, Stanford, California
  - Pfizer Investigational Site, Boulder, Colorado
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Danbury, Connecticut
  - Pfizer Investigational Site, Hamden, Connecticut
  - Pfizer Investigational Site, Trumbull, Connecticut
  - Pfizer Investigational Site, New Port Richey, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Plantation, Florida
  - Pfizer Investigational Site, Port Richey, Florida
  - Pfizer Investigational Site, Tamarac, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Marietta, Georgia
  - Pfizer Investigational Site, Maywood, Illinois
  - Pfizer Investigational Site, Oakbrook Terrace, Illinois
  - Pfizer Investigational Site, Rockford, Illinois
  - Pfizer Investigational Site, Springfield, Illinois
  - Pfizer Investigational Site, Vernon Hills, Illinois
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Leominster, Massachusetts
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, Edina, Minnesota
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Orchard Park, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Asheville, North Carolina
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Bethlehem, Pennsylvania
  - Pfizer Investigational Site, Wyomissing, Pennsylvania
  - Pfizer Investigational Site, Greenville, South Carolina
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Tacoma, Washington
  - Pfizer Investigational Site, Clarksburg, West Virginia
- Australia (6):
  - Pfizer Investigational Site, Campsie, New South Wales
  - Pfizer Investigational Site, Cairns, Queensland
  - Pfizer Investigational Site, Maroochydore, Queensland
  - Pfizer Investigational Site, Woodville, South Australia
  - Pfizer Investigational Site, Malvern East, Victoria
  - Pfizer Investigational Site, Shenton Park, Western Australia
- Chile (4):
  - Pfizer Investigational Site, Viña del Mar, Región de Valparaíso
  - Pfizer Investigational Site, Santiago, RM
  - Pfizer Investigational Site, Providencia, Santiago, RM
  - Pfizer Investigational Site, Viña del Mar
- China (14):
  - Pfizer Investigational Site, Hefei, Anhui
  - Pfizer Investigational Site, Guangzhou, Guangdong
  - Pfizer Investigational Site, Wuhan, Hubei
  - Pfizer Investigational Site, Changsha, Hunan
  - Pfizer Investigational Site, Nanjing, Jiangsu
  - Pfizer Investigational Site, Suzhou, Jiangsu
  - Pfizer Investigational Site, Jinan, Shandong
  - Pfizer Investigational Site, Qingdao, Shandong
  - Pfizer Investigational Site, Xi’an, Shanxi
  - Pfizer Investigational Site, Chengdu, Sichuan
  - Pfizer Investigational Site, Hangzhou, Zhejiang
  - Pfizer Investigational Site, Beijing
  - Pfizer Investigational Site, Shanghai
  - Pfizer Investigational Site, Tianjin
- Colombia (3):
  - Pfizer Investigational Site, Barranquilla, Atlántico
  - Pfizer Investigational Site, Bogota, Cundinamarca
  - Pfizer Investigational Site, Bucaramanga, Santander Department
- Croatia (2):
  - Pfizer Investigational Site, Opatija
  - Pfizer Investigational Site, Zagreb
- Pfizer Investigational Site, Frederiksberg, Denmark
- Finland (3):
  - Pfizer Investigational Site, Helsinki
  - Pfizer Investigational Site, Hyvinkää
  - Pfizer Investigational Site, Tampere
- Germany (6):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Dresden
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, Nuremberg
  - Pfizer Investigational Site, Rheine
- Pfizer Investigational Site, Maroussi Athens, Greece
- Malaysia (4):
  - Pfizer Investigational Site, Putrajaya, Kuala Lumpur
  - Pfizer Investigational Site, Seremban, Negeri Sembilan
  - Pfizer Investigational Site, Batu Caves, Selangor
  - Pfizer Investigational Site, Subang Jaya, Selangor
- Mexico (5):
  - Pfizer Investigational Site, Torreón, Coahuila
  - Pfizer Investigational Site, Morelia, Michoacán
  - Pfizer Investigational Site, Cuernavaca, Morelos
  - Pfizer Investigational Site, México, Querétaro
  - Pfizer Investigational Site, Mérida, Yucatán
- Poland (4):
  - Pfizer Investigational Site, Bialystok
  - Pfizer Investigational Site, Kościan
  - Pfizer Investigational Site, Poznan
  - Pfizer Investigational Site, Torun
- Russia (2):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Petrozavodsk
- Slovakia (6):
  - Pfizer Investigational Site, Nové Zámky
  - Pfizer Investigational Site, Poprad
  - Pfizer Investigational Site, Považská Bystrica
  - Pfizer Investigational Site, Rimavská Sobota
  - Pfizer Investigational Site, Senica
  - Pfizer Investigational Site, Žilina
- Spain (5):
  - Pfizer Investigational Site, A Coruña, A Coruña
  - Pfizer Investigational Site, Santiago de Compostela, A Coruña
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Málaga, Malaga
  - Pfizer Investigational Site, Seville, Sevilla
- Sweden (3):
  - Pfizer Investigational Site, Falun
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Uppsala
- Thailand (3):
  - Pfizer Investigational Site, Rajathevee, Bangkok
  - Pfizer Investigational Site, Amphoe Muang, Chiang Mai
  - Pfizer Investigational Site, Muang District, Khonkaen
- United Kingdom (4):
  - Pfizer Investigational Site, Metropolitan Borough of Wirral, Merseyside
  - Pfizer Investigational Site, Cannock, Staffs
  - Pfizer Investigational Site, Solihull, West Midlands
  - Pfizer Investigational Site, Newcastle upon Tyne
- Venezuela (2):
  - Pfizer Investigational Site, Caracas, DC/ Municipio Libertados
  - Pfizer Investigational Site, Caracas, Distrito Federal

REFERENCES:
- [Derived] Strand V, Schulze-Koops H, Al-Emadi S, Kinch CD, Gruben D, Germino R, Connell CA, Mysler E. Sex differences in the efficacy, safety and persistence of tofacitinib in patients with rheumatoid arthritis: a post hoc analysis of phase III and long-term extension trials. BMJ Open. 2025 Dec 24;15(12):e082366. doi: 10.1136/bmjopen-2023-082366. PMID 41448717
- [Derived] Hetland ML, Strangfeld A, Bonfanti G, Soudis D, Deuring JJ, Edwards RA. Machine learning prediction and explanatory models of serious infections in patients with rheumatoid arthritis treated with tofacitinib. Arthritis Res Ther. 2024 Aug 27;26(1):153. doi: 10.1186/s13075-024-03376-9. PMID 39192350
- [Derived] Wright GC, Mysler E, Kwok K, Cadatal MJ, Germino R, Yndestad A, Kinch CD, Ogdie A. Impact of Race on the Efficacy and Safety of Tofacitinib in Rheumatoid Arthritis: Post Hoc Analysis of Pooled Clinical Trials. Rheumatol Ther. 2024 Oct;11(5):1135-1164. doi: 10.1007/s40744-024-00677-y. Epub 2024 Jul 3. PMID 38958913
- [Derived] Citera G, Jain R, Irazoque F, Madariaga H, Gruben D, Wang L, Stockert L, Santana K, Ebrahim A, Ponce de Leon D. Tofacitinib Efficacy in Patients with Rheumatoid Arthritis and Probable Depression/Anxiety: Post Hoc Analysis of Phase 3 and 3b/4 Randomized Controlled Trials. Rheumatol Ther. 2024 Feb;11(1):35-50. doi: 10.1007/s40744-023-00612-7. Epub 2023 Nov 5. PMID 37925660
- [Derived] Tesser J, Gul A, Olech E, Oelke K, Lukic T, Kwok K, Ebrahim A. Efficacy and safety of tofacitinib in patients with rheumatoid arthritis by previous treatment: post hoc analysis of phase II/III trials. Arthritis Res Ther. 2023 Nov 2;25(1):214. doi: 10.1186/s13075-023-03154-z. PMID 37919780
- [Derived] Charles-Schoeman C, Hyde C, Guan S, Parikh N, Wang J, Shahbazian A, Stockert L, Andrews J. Relationship Between Paraoxonase-1 Genotype and Activity, and Major Adverse Cardiovascular Events and Malignancies in Patients With Rheumatoid Arthritis Receiving Tofacitinib. J Rheumatol. 2023 Jul 15:jrheum.2023-0112. doi: 10.3899/jrheum.2023-0112. Online ahead of print. PMID 37453736
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Dougados M, Taylor PC, Bingham CO 3rd, Fallon L, Brault Y, Roychoudhury S, Wang L, Kessouri M. The effect of tofacitinib on residual pain in patients with rheumatoid arthritis and psoriatic arthritis. RMD Open. 2022 Sep;8(2):e002478. doi: 10.1136/rmdopen-2022-002478. PMID 36814062
- [Derived] Hansen KE, Mortezavi M, Nagy E, Wang C, Connell CA, Radi Z, Litman HJ, Adami G, Rossini M. Fracture in clinical studies of tofacitinib in rheumatoid arthritis. Ther Adv Musculoskelet Dis. 2022 Dec 27;14:1759720X221142346. doi: 10.1177/1759720X221142346. eCollection 2022. PMID 36601090
- [Derived] Curtis JR, Yamaoka K, Chen YH, Bhatt DL, Gunay LM, Sugiyama N, Connell CA, Wang C, Wu J, Menon S, Vranic I, Gomez-Reino JJ. Malignancy risk with tofacitinib versus TNF inhibitors in rheumatoid arthritis: results from the open-label, randomised controlled ORAL Surveillance trial. Ann Rheum Dis. 2023 Mar;82(3):331-343. doi: 10.1136/ard-2022-222543. Epub 2022 Dec 5. PMID 36600185
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Dikranian AH, Gonzalez-Gay MA, Wellborne F, Alvaro-Gracia JM, Takiya L, Stockert L, Paulissen J, Shi H, Tatulych S, Curtis JR. Efficacy of tofacitinib in patients with rheumatoid arthritis stratified by baseline body mass index: an analysis of pooled data from phase 3 studies. RMD Open. 2022 May;8(1):e002103. doi: 10.1136/rmdopen-2021-002103. PMID 35577477
- [Derived] Bartlett SJ, Bingham CO, van Vollenhoven R, Murray C, Gruben D, Gold DA, Cella D. The impact of tofacitinib on fatigue, sleep, and health-related quality of life in patients with rheumatoid arthritis: a post hoc analysis of data from Phase 3 trials. Arthritis Res Ther. 2022 Apr 5;24(1):83. doi: 10.1186/s13075-022-02724-x. PMID 35382883
- [Derived] Dikranian A, Gold D, Bessette L, Nash P, Azevedo VF, Wang L, Woolcott J, Shapiro AB, Szumski A, Fleishaker D, Wollenhaupt J. Frequency and Duration of Early Non-serious Adverse Events in Patients with Rheumatoid Arthritis and Psoriatic Arthritis Treated with Tofacitinib. Rheumatol Ther. 2022 Apr;9(2):411-433. doi: 10.1007/s40744-021-00405-w. Epub 2021 Dec 17. PMID 34921355
- [Derived] Winthrop KL, Curtis JR, Yamaoka K, Lee EB, Hirose T, Rivas JL, Kwok K, Burmester GR. Clinical Management of Herpes Zoster in Patients With Rheumatoid Arthritis or Psoriatic Arthritis Receiving Tofacitinib Treatment. Rheumatol Ther. 2022 Feb;9(1):243-263. doi: 10.1007/s40744-021-00390-0. Epub 2021 Dec 6. PMID 34870800
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Wang L, Chen C, Kwok K, Biswas P, Shapiro A, Madsen A, Wollenhaupt J. Long-term safety of tofacitinib up to 9.5 years: a comprehensive integrated analysis of the rheumatoid arthritis clinical development programme. RMD Open. 2020 Oct;6(3):e001395. doi: 10.1136/rmdopen-2020-001395. PMID 33127856
- [Derived] Strand V, Kaine J, Alten R, Wallenstein G, Diehl A, Shi H, Germino R, Murray CW. Associations between Patient Global Assessment scores and pain, physical function, and fatigue in rheumatoid arthritis: a post hoc analysis of data from phase 3 trials of tofacitinib. Arthritis Res Ther. 2020 Oct 15;22(1):243. doi: 10.1186/s13075-020-02324-7. PMID 33059710
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Li ZG, Liu Y, Xu HJ, Chen ZW, Bao CD, Gu JR, Zhao DB, An Y, Hwang LJ, Wang L, Kremer J, Wu QZ. Efficacy and Safety of Tofacitinib in Chinese Patients with Rheumatoid Arthritis. Chin Med J (Engl). 2018 Nov 20;131(22):2683-2692. doi: 10.4103/0366-6999.245157. PMID 30425195
- [Derived] Kivitz AJ, Cohen S, Keystone E, van Vollenhoven RF, Haraoui B, Kaine J, Fan H, Connell CA, Bananis E, Takiya L, Fleischmann R. A pooled analysis of the safety of tofacitinib as monotherapy or in combination with background conventional synthetic disease-modifying antirheumatic drugs in a Phase 3 rheumatoid arthritis population. Semin Arthritis Rheum. 2018 Dec;48(3):406-415. doi: 10.1016/j.semarthrit.2018.07.006. Epub 2018 Jul 19. PMID 30177460
- [Derived] Hall S, Nash P, Rischmueller M, Bossingham D, Bird P, Cook N, Witcombe D, Soma K, Kwok K, Thirunavukkarasu K. Tofacitinib, an Oral Janus Kinase Inhibitor: Pooled Efficacy and Safety Analyses in an Australian Rheumatoid Arthritis Population. Rheumatol Ther. 2018 Dec;5(2):383-401. doi: 10.1007/s40744-018-0118-2. Epub 2018 Jun 11. PMID 29949132
- [Derived] Bird P, Bensen W, El-Zorkany B, Kaine J, Manapat-Reyes BH, Pascual-Ramos V, Witcombe D, Soma K, Zhang R, Thirunavukkarasu K. Tofacitinib 5 mg Twice Daily in Patients with Rheumatoid Arthritis and Inadequate Response to Disease-Modifying Antirheumatic Drugs: A Comprehensive Review of Phase 3 Efficacy and Safety. J Clin Rheumatol. 2019 Apr;25(3):115-126. doi: 10.1097/RHU.0000000000000786. PMID 29794874
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Thirunavukkarasu K, DeMasi R, Geier J, Kwok K, Wang L, Riese R, Wollenhaupt J. Long-term safety of tofacitinib for the treatment of rheumatoid arthritis up to 8.5 years: integrated analysis of data from the global clinical trials. Ann Rheum Dis. 2017 Jul;76(7):1253-1262. doi: 10.1136/annrheumdis-2016-210457. Epub 2017 Jan 31. PMID 28143815
- [Derived] Strand V, Kremer JM, Gruben D, Krishnaswami S, Zwillich SH, Wallenstein GV. Tofacitinib in Combination With Conventional Disease-Modifying Antirheumatic Drugs in Patients With Active Rheumatoid Arthritis: Patient-Reported Outcomes From a Phase III Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2017 Apr;69(4):592-598. doi: 10.1002/acr.23004. PMID 27565000
- [Derived] Charles-Schoeman C, Burmester G, Nash P, Zerbini CA, Soma K, Kwok K, Hendrikx T, Bananis E, Fleischmann R. Efficacy and safety of tofacitinib following inadequate response to conventional synthetic or biological disease-modifying antirheumatic drugs. Ann Rheum Dis. 2016 Jul;75(7):1293-301. doi: 10.1136/annrheumdis-2014-207178. Epub 2015 Aug 14. PMID 26275429
- [Derived] Cohen S, Radominski SC, Gomez-Reino JJ, Wang L, Krishnaswami S, Wood SP, Soma K, Nduaka CI, Kwok K, Valdez H, Benda B, Riese R. Analysis of infections and all-cause mortality in phase II, phase III, and long-term extension studies of tofacitinib in patients with rheumatoid arthritis. Arthritis Rheumatol. 2014 Nov;66(11):2924-37. doi: 10.1002/art.38779. PMID 25047021
- [Derived] Kremer J, Li ZG, Hall S, Fleischmann R, Genovese M, Martin-Mola E, Isaacs JD, Gruben D, Wallenstein G, Krishnaswami S, Zwillich SH, Koncz T, Riese R, Bradley J. Tofacitinib in combination with nonbiologic disease-modifying antirheumatic drugs in patients with active rheumatoid arthritis: a randomized trial. Ann Intern Med. 2013 Aug 20;159(4):253-61. doi: 10.7326/0003-4819-159-4-201308200-00006. PMID 24026258
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921046&StudyName=A%20Study%20Comparing%202%20Doses%20Of%20CP-690%2C550%20Vs.%20Placebo%20For%20The%20Treatment%20Of%20Rheumatoid%20Arthritis%20In%20Patients%20On%20Other%20Background%20Arthri

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-690,550 5 mg: CP-690,550 5 milligram (mg) tablet orally twice daily up to Month 12.
- CP-690,550 10 mg: CP-690,550 10 mg tablet orally twice daily up to Month 12.
- Placebo Then CP-690,550 5 mg: Placebo matched to CP-690,550 tablet orally twice daily for 3 to 6 months. Response was assessed at Month 3 and participants who failed to achieve at least 20 percent (%) reduction in both swollen and tender joint counts from baseline, received CP-690,550 5 mg tablet orally twice daily up to Month 12. At Month 6, remaining participants received CP-690,550 5 mg tablet orally twice daily up to Month 12.
- Placebo Then CP-690,550 10 mg: Placebo matched to CP-690,550 tablet orally twice daily for 3 to 6 months. Response was assessed at Month 3 and participants who failed to achieve at least 20 percent (%) reduction in both swollen and tender joint counts from baseline, received CP-690,550 10 mg tablet orally twice daily up to Month 12. At Month 6, remaining participants received CP-690,550 10 mg tablet orally twice daily up to Month 12.
Period: Overall Study
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo Then CP-690,550 5 mg | Placebo Then CP-690,550 10 mg
Started | 318 | 318 | 79 | 80
Treated | 315 | 318 | 79 | 80
Completed | 261 | 252 | 71 | 67
Not Completed | 57 | 66 | 8 | 13
Not completed — Randomized but not treated | 3 | 0 | 0 | 0
Not completed — Death | 0 | 2 | 0 | 0
Not completed — Adverse Event | 20 | 29 | 2 | 3
Not completed — Lack of Efficacy | 16 | 12 | 3 | 3
Not completed — Other | 9 | 16 | 1 | 6
Not completed — Lost to Follow-up | 1 | 2 | 2 | 0
Not completed — Withdrawal by Subject | 8 | 5 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo Then CP-690,550 5 mg | Placebo Then CP-690,550 10 mg | Total
Number analyzed (Participants) | 315 | 318 | 79 | 80 | 792
Age Continuous [Mean (Standard Deviation); unit: Years] | 52.7 (11.7) | 51.9 (11.8) | 50.8 (11.2) | 53.3 (10.8) | 52.3 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 264 | 258 | 63 | 60 | 645
  Male | 51 | 60 | 16 | 20 | 147

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response at Month 6
Description: ACR20 response: greater than or equal to (>=) 20 percent (%) improvement in tender joint count (TJC); >= 20% improvement in swollen joint count (SJC); and >= 20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP). For comparison of CP-690,550 with placebo, placebo sequences were combined into single reporting group for Month 6 analysis.
Time Frame: Month 6
Population: Full analysis set (FAS) population included all randomized participants who received at least 1 dose of study medication. N (number of participants analyzed)=participants who were evaluable for this measure. Missing values due to withdrawal, advancement to active treatment before Month 6 were imputed using non-responder imputation (NRI) method.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Placebo matched to CP-690,550 tablet orally twice daily for 3 to 6 months. Response was assessed at Month 3 and participants who failed to achieve at least 20% reduction in both swollen and tender joint counts from baseline, received CP-690,550 5 mg or 10 mg tablet orally twice daily up to Month 12. At Month 6, remaining participants received CP-690,550 5 mg or 10 mg tablet orally twice daily up to Month 12.
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 311 | 309 | 157
percentage of participants | 52.73 | 58.25 | 31.21
Statistical Analysis 1: Comparison: CP-690,550 10 mg vs Placebo; Normal approximation to the binomial distribution was used to test the superiority of each dose of CP-690,550 10 mg to placebo and 2-sided 95% confidence interval (CI) was evaluated for the difference in percentages; Test type: Superiority or Other; p < 0.0001, Normal approximation — A step-down procedure was used to control for multiple comparisons. In order for the comparison to 5 mg to be statistically significant, the comparison to 10 mg had to be statistically significant; Percent difference = 27.04, 95% CI 2-sided [17.94 to 36.13]
Statistical Analysis 2: Comparison: CP-690,550 5 mg vs Placebo; Normal approximation to the binomial distribution was used to test the superiority of each dose of CP-690,550 5 mg to placebo and 2-sided 95% CI was evaluated for the difference in percentages; Test type: Superiority or Other; p < 0.0001, Normal Approximation — [p-value comment as in outcome 1, analysis 1]; Percent Difference = 21.52, 95% CI 2-sided [12.39 to 30.65]

2. Primary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Month 3
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities:dress/groom;arise;eat; walk;reach;grip; hygiene;common activities over past week. Each item scored on 4-point scale from 0-3:0=no difficulty;1=some difficulty;2=much difficulty;3=unable to do. Overall score was computed as sum of domain scores and divided by number of domains answered. Total possible score range 0-3:0=least difficulty and 3=extreme difficulty. For comparison of CP-690,550 with placebo, placebo sequences were combined into single reporting group for Month 3 analysis.
Time Frame: Baseline, Month 3
Population: FAS population included all randomized participants who received at least 1 dose of study medication. N (number of participants analyzed)=participants who were evaluable for this measure. Here 'n' is number of participants evaluable at specific time points for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Placebo matched to CP-690,550 tablet orally twice daily for 3 to 6 months. Response was assessed at Month 3 and participants who failed to achieve at least 20 percent (%) reduction in both swollen and tender joint counts from baseline, received CP-690,550 5 mg or 10 mg tablet orally twice daily up to Month 12. At Month 6, remaining participants received CP-690,550 5 mg or 10 mg tablet orally twice daily up to Month 12.
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 311 | 315 | 157
units on a scale
  Baseline (n= 311, 315, 157) | 1.44 (0.69) | 1.43 (0.68) | 1.35 (0.66)
  Change at Month 3 (n= 292, 292, 147) | -0.45 (0.53) | -0.54 (0.60) | -0.16 (0.54)
Statistical Analysis 1: Comparison: CP-690,550 10 mg vs Placebo; Least squares mean difference (LS Mean Difference) and corresponding 95% CI was calculated using a mixed effect repeated measure model with treatments, visits and treatment-by-visit interaction as fixed effects and participants as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — A step-down procedure was used to control for multiple comparisons. For the comparison of 10 mg to placebo to be statistically significant, the comparison of 10 mg to placebo in ACR20 had to be significant; LS mean difference = -0.35, 95% CI 2-sided [-0.44 to -0.26], Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: CP-690,550 5 mg vs Placebo; LS Mean Difference and corresponding 95% CI was calculated using a mixed effect repeated measure model with treatments, visits and treatment-by-visit interaction as fixed effects and participants as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — A step-down procedure was used to control for multiple comparisons. For comparison of 5 mg to placebo to be statistically significant, comparison of 10 mg to placebo and comparison of 5 mg to placebo in ACR20 had to be statistically significant; LS mean difference = -0.26, 95% CI 2-sided [-0.35 to -0.16], Standard Error of Mean 0.05

3. Primary Outcome: Percentage of Participants Achieving Disease Activity Score Using 28-Joint Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR])Less Than 2.6 at Month 6
Description: DAS28-4 (ESR) was calculated from SJC and TJC using 28 joints count, erythrocyte sedimentation rate (ESR) (millimeters/hour[mm/hour]) and patient's global assessment (PtGA) of disease activity(participant rated arthritis activity assessment). Total score range:0-9.4, higher score=more disease activity. DAS28-4 (ESR) less than or equal to (<=)3.2 implied low disease activity, greater than (>)3.2 to 5.1 implied moderate to high disease activity, less than (<)2.6=remission. For comparison of CP-690,550 with placebo, placebo sequences were combined into single reporting group for Month 6 analysis.
Time Frame: Month 6
Population: FAS population included all randomized participants who received at least 1 dose of study medication. N (number of participants analyzed) signifies those participants who were evaluable for this measure. Missing values due to withdrawal, advancement to active treatment before Month 6 were imputed using NRI method.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 263 | 270 | 148
percentage of participants | 9.13 | 13.33 | 2.70
Statistical Analysis 1: Comparison: CP-690,550 10 mg vs Placebo; Normal approximation to the binomial distribution was used to test the superiority of each dose of CP-690,550 10 mg to placebo and 2-sided 95% CI was evaluated for the difference in percentages; Test type: Superiority or Other; p < 0.0001, Normal Approximation — A step-down procedure was used to control for multiple comparisons. For the comparison of 10 mg to placebo to be statistically significant, the comparison of 10 mg to placebo in HAQ-DI had to be significant; Percent difference = 10.63, 95% CI 2-sided [5.80 to 15.45]
Statistical Analysis 2: Comparison: CP-690,550 5 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0038, Normal Approximation — A step-down procedure was used to control for multiple comparisons. For comparison of 5 mg to placebo to be statistically significant, comparison of 10 mg to placebo and comparison of 5 mg to placebo in HAQ-DI had to be statistically significant; Percent difference = 6.42, 95% CI 2-sided [2.07 to 10.77]

4. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) at Week 2, Month 1, 2, 3, 4.5 and 6
Description: ACR20 response: >=20% improvement in tender joint count; >=20% improvement in swollen joint count; and >=20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of HAQ); and CRP.
Time Frame: Week 2, Month 1, 2, 3, 4.5, 6
Population: FAS population. N (number of participants analyzed)=participants who were evaluable for this measure. Missing values due to withdrawal from study or advancement to active treatment, before Month 6 was imputed using NRI method.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 311 | 309 | 157
percentage of participants
  Week 2 | 27.33 | 32.25 | 10.90
  Month 1 | 38.59 | 48.54 | 22.93
  Month 2 | 54.02 | 64.40 | 26.11
  Month 3 | 56.27 | 64.72 | 27.39
  Month 4.5 | 50.80 | 57.93 | 25.48
  Month 6 | 52.73 | 58.25 | 31.21

5. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) at Month 9 and 12
Description: as for outcome 4
Time Frame: Month 9, 12
Population: FAS population. 'N' (number of participants analyzed)=participants who were evaluable for this measure. Missing values due to withdrawal from study or advancement to active treatment, before Month 6 was imputed using NRI method.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo Then CP-690,550 5 mg | Placebo Then CP-690,550 10 mg
Number analyzed (Participants) | 311 | 309 | 79 | 78
percentage of participants
  Month 9 | 50.48 | 62.14 | 37.97 | 34.62
  Month 12 | 51.45 | 56.63 | 31.65 | 34.62

6. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) at Week 2, Month 1, 2, 3, 4.5 and 6
Description: ACR50 response: >=50% improvement in tender joint count; >=50% improvement in swollen joint count; and >=50% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of HAQ); and CRP.
Time Frame: Week 2, Month 1, 2, 3, 4.5, 6
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 311 | 309 | 157
percentage of participants
  Week 2 | 5.79 | 8.14 | 1.28
  Month 1 | 11.58 | 18.12 | 1.27
  Month 2 | 23.15 | 29.77 | 4.46
  Month 3 | 27.33 | 33.98 | 9.55
  Month 4.5 | 27.97 | 33.33 | 8.28
  Month 6 | 33.76 | 36.57 | 12.74

7. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) at Month 9 and 12
Description: as for outcome 6
Time Frame: Month 9, 12
Population: FAS population included participants who received at least 1 dose of study medication. 'N' (number of participants analyzed)signifies those participants who were evaluable for this measure. Missing values due to withdrawal, advancement to active treatment before Month 6 were imputed using NRI method.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo Then CP-690,550 5 mg | Placebo Then CP-690,550 10 mg
Number analyzed (Participants) | 311 | 309 | 79 | 78
percentage of participants
  Month 9 | 31.51 | 43.04 | 25.32 | 26.92
  Month 12 | 33.44 | 42.72 | 24.05 | 25.64

8. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) at Week 2, Month 1, 2, 3, 4.5 and 6
Description: ACR70 response: >=70% improvement in tender joint count; >=70% improvement in swollen joint count; and >=70% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of HAQ); and CRP.
Time Frame: Week 2, Month 1, 2, 3, 4.5, 6
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 311 | 309 | 157
percentage of participants
  Week 2 | 0.32 | 2.28 | 0.00
  Month 1 | 3.54 | 7.12 | 0.00
  Month 2 | 9.00 | 10.36 | 1.27
  Month 3 | 8.36 | 14.24 | 1.91
  Month 4.5 | 11.90 | 18.12 | 3.18
  Month 6 | 13.18 | 16.18 | 3.18

9. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) at Month 9 and 12
Description: as for outcome 8
Time Frame: Month 9, 12
Population: FAS population included participants who received at least 1 dose of study medication. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. Missing values due to withdrawal, advancement to active treatment before Month 6 were imputed using NRI method.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo Then CP-690,550 5 mg | Placebo Then CP-690,550 10 mg
Number analyzed (Participants) | 311 | 309 | 79 | 78
percentage of participants
  Month 9 | 14.15 | 25.24 | 10.13 | 11.54
  Month 12 | 19.29 | 25.57 | 13.92 | 20.51

10. Secondary Outcome: Disease Activity Score Using 28-Joint Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP]) at Baseline, Week 2, Month 1, 2, 3, 4.5 and 6
Description: DAS28-3 (CRP) was calculated from SJC and TJC using 28 joint count and CRP (mg/L). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3 (CRP) =<3.2 implied low disease activity, >3.2 to 5.1 implied moderate to high disease activity and <2.6 implied remission.
Time Frame: Week 2, Month 1, 2, 3, 4.5, 6
Population: FAS population included participants who received at least 1 dose of study medication. 'n' signifies those participants who were evaluable for this measure at given time points for each group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 312 | 315 | 158
units on a scale
  Baseline (n=312, 315, 158) | 5.21 (0.92) | 5.26 (0.96) | 5.22 (0.92)
  Week 2 (n=309, 304, 156) | 4.41 (1.10) | 4.18 (1.09) | 4.92 (1.01)
  Month 1 (n=304, 300, 151) | 4.08 (1.13) | 3.83 (1.12) | 4.68 (1.09)
  Month 2 (n=294, 300, 148) | 3.70 (1.20) | 3.49 (1.15) | 4.59 (1.16)
  Month 3 (n=293, 291, 147) | 3.62 (1.22) | 3.44 (1.15) | 4.51 (1.15)
  Month 4.5 (n=281,286,71) | 3.46 (1.27) | 3.15 (1.12) | 3.92 (1.18)
  Month 6 (n=279,278,68) | 3.39 (1.21) | 3.09 (1.13) | 3.60 (1.12)

11. Secondary Outcome: Disease Activity Score Using 28-Joint Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP]) at Month 9 and 12
Description: as for outcome 10
Time Frame: Month 9, 12
Population: FAS population included participants who received at least 1 dose of study medication. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo Then CP-690,550 5 mg | Placebo Then CP-690,550 10 mg
Number analyzed (Participants) | 267 | 263 | 72 | 68
units on a scale
  Month 9 | 3.21 (1.14) | 2.88 (1.05) | 3.22 (1.05) | 2.83 (0.93)
  Month 12 | 3.08 (1.19) | 2.81 (1.04) | 3.03 (1.15) | 2.99 (1.06)

12. Secondary Outcome: Disease Activity Score Using 28-Joint Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR]) at Baseline, Month 3 and 6
Description: DAS28-4 (ESR) calculated from SJC and TJC using 28 joint count, ESR (mm/hour) and PGA of disease activity (participant rated arthritis activity assessment with transformed score ranging 0 to 10; higher score indicated greater affectation due to disease activity). Total score range:0 to 9.4, higher score indicated more disease activity. DAS28-4 (ESR) =<3.2 implied low disease activity, >3.2 to 5.1 implied moderate to high disease activity and <2.6 implied remission.
Time Frame: Baseline, Month 3, 6
Population: FAS population included participants who received at least 1 dose of study medication. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n' signifies those participants who were evaluable for this measure at given time points for each group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 309 | 313 | 158
units on a scale
  Baseline (n=309,313,158) | 6.29 (0.96) | 6.36 (1.01) | 6.30 (0.92)
  Month 3 (n=206,263,140) | 4.41 (1.39) | 4.20 (1.30) | 5.32 (1.26)
  Month 6 (n=241,248,62) | 4.14 (1.34) | 3.84 (1.26) | 4.34 (1.19)

13. Secondary Outcome: Disease Activity Score Using 28-Joint Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR]) at Month 12
Description: as for outcome 12
Time Frame: Month 12
Population: FAS population included participants who received at least 1 dose of study medication. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo Then CP-690,550 5 mg | Placebo Then CP-690,550 10 mg
Number analyzed (Participants) | 220 | 226 | 63 | 62
units on a scale | 3.82 (1.30) | 3.50 (1.11) | 3.76 (1.31) | 3.62 (1.19)

14. Secondary Outcome: Disease Activity Score Using 28-Joint Count and C-Reactive Protein (4 Variables) (DAS28-4 [CRP])
Description: DAS28-4 (CRP) was calculated from SJC and TJC using the 28 joints count, CRP [mg/L] and PtGA of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-4 [CRP] <=3.2 implied low disease activity, DAS28-4 [CRP] >3.2 to 5.1 implied moderate to high disease activity and DAS28 <2.6 implied remission.
Time Frame: Baseline, Week 2, Month 1, 2, 3, 4.5, 6, 9, 12
Population: Since DAS28-4 (CRP) was determined to provide no new information over DAS28-4 (ESR) and DAS28-3 (CRP), there was a change in planned analysis and data was not analyzed for DAS28-4 (CRP).
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo Then CP-690,550 5 mg | Placebo Then CP-690,550 10 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Secondary Outcome: Disease Activity Score Using 28-Joint Count and Erythrocyte Sedimentation Rate (3 Variables) (DAS28-3 [ESR])
Description: DAS28-3 (ESR) was calculated from the number of SJC and TJC using the 28 joints count and ESR (mm/hr). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3 (ESR) <=3.2 implied low disease activity, >3.2 to 5.1 implied moderate to high disease activity and <2.6 implied remission.
Time Frame: Baseline, Month 3, 6, 12
Population: Since DAS28-3 (ESR) was determined to provide no new information over DAS28-4 (ESR) and DAS28-3 (CRP), there was a change in planned analysis and data was not analyzed for DAS28-3 (ESR).
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo Then CP-690,550 5 mg | Placebo Then CP-690,550 10 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

16. Secondary Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI) at Baseline, Week 2, Month 1, 2, 3, 4.5 and 6
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0=least difficulty and 3=extreme difficulty.
Time Frame: Baseline, Week 2, Month 1, 2, 3, 4.5, 6
Population: FAS population. N (number of participants analyzed)=participants who were evaluable for this measure. 'n'=participants evaluable at given time point for each group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 311 | 315 | 157
units on a scale
  Baseline (n = 311, 315, 157) | 1.44 (0.69) | 1.43 (0.68) | 1.35 (0.66)
  Week 2 (n = 310, 305, 156) | 1.24 (0.69) | 1.14 (0.67) | 1.28 (0.66)
  Month 1 (n = 304, 303, 154) | 1.12 (0.67) | 1.01 (0.65) | 1.20 (0.67)
  Month 2 (n = 299, 300, 150) | 1.03 (0.68) | 0.93 (0.66) | 1.20 (0.63)
  Month 3 (n = 293, 292, 148) | 0.98 (0.67) | 0.88 (0.67) | 1.16 (0.67)
  Month 4.5 (n = 282, 289, 71) | 0.97 (0.68) | 0.84 (0.67) | 0.95 (0.62)
  Month 6 (n = 278, 279, 68) | 0.91 (0.67) | 0.81 (0.65) | 0.93 (0.61)

17. Secondary Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI) at Month 9 and 12
Description: as for outcome 16
Time Frame: Month 9, Month 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo Then CP-690,550 5 mg | Placebo Then CP-690,550 10 mg
Number analyzed (Participants) | 266 | 264 | 72 | 70
units on a scale
  Month 9 | 0.89 (0.68) | 0.71 (0.64) | 0.85 (0.65) | 0.70 (0.64)
  Month 12 | 0.86 (0.68) | 0.73 (0.64) | 0.81 (0.68) | 0.73 (0.69)

18. Secondary Outcome: Patient Assessment of Arthritis Pain at Baseline, Week 2, Month 1, 2, 3, 4.5 and 6
Description: Participants rated the severity of arthritis pain on a 0 to 100 millimeter (mm) visual analogue scale (VAS), where 0 mm = no pain and 100 mm = most severe pain.
Time Frame: Baseline, Week 2, Month 1, 2, 3, 4.5, 6
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 311 | 315 | 158
mm
  Baseline (n = 311, 315, 158) | 57.08 (23.82) | 58.58 (22.19) | 57.11 (22.84)
  Week 2 (n = 310, 306, 156) | 46.81 (22.82) | 41.85 (22.49) | 51.01 (24.45)
  Month 1 (n = 304, 303, 154) | 40.17 (23.20) | 37.08 (22.14) | 45.69 (25.00)
  Month 2 (n = 299, 301, 150) | 36.40 (22.63) | 32.84 (21.71) | 47.30 (24.29)
  Month 3 (n = 294, 292, 148) | 34.92 (23.03) | 32.96 (23.10) | 46.59 (27.14)
  Month 4.5 (n = 284, 289, 71) | 34.43 (22.68) | 32.62 (21.74) | 40.23 (24.44)
  Month 6 (n = 279, 280, 68) | 31.07 (21.84) | 29.94 (21.53) | 34.19 (21.69)

19. Secondary Outcome: Patient Assessment of Arthritis Pain at Month 9 and 12
Description: Participants rated the severity of arthritis pain on a 0 to 100 mm VAS, where 0 mm = no pain and 100 mm = most severe pain.
Time Frame: Month 9, 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo Then CP-690,550 5 mg | Placebo Then CP-690,550 10 mg
Number analyzed (Participants) | 267 | 264 | 72 | 70
mm
  Month 9 | 30.78 (22.28) | 27.13 (20.77) | 29.50 (21.34) | 25.26 (21.96)
  Month 12 | 30.18 (23.11) | 25.43 (20.57) | 28.20 (22.46) | 25.39 (22.71)

20. Secondary Outcome: Patient Global Assessment (PtGA) of Arthritis Pain at Baseline, Week 2, Month 1, 2, 3, 4.5 and 6
Description: Participants answered: "Considering all the ways your arthritis affects you, how are you feeling today?" Participants responded by using a 0 - 100 mm VAS where 0 = very well and 100 = very poorly.
Time Frame: Baseline, Week 2, Month 1, 2, 3, 4.5, 6
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 311 | 315 | 158
mm
  Baseline (n=311,315,158) | 59.03 (22.89) | 60.22 (22.53) | 57.92 (23.33)
  Week 2 (n=310,306,156) | 46.59 (22.52) | 42.99 (22.16) | 51.27 (23.97)
  Month 1 (n=303,303,154) | 40.50 (23.29) | 36.53 (21.42) | 46.25 (24.22)
  Month 2 (n=299,301,150) | 37.18 (22.52) | 33.80 (22.21) | 50.42 (23.56)
  Month 3 (n=294,292,148) | 36.27 (22.64) | 33.43 (22.55) | 47.09 (26.13)
  Month 4.5 (n=284,289,71) | 35.92 (22.69) | 34.05 (22.09) | 41.03 (23.75)
  Month 6 (n=279,280,68) | 33.75 (23.01) | 31.31 (21.55) | 35.47 (20.28)

21. Secondary Outcome: Patient Global Assessment (PtGA) of Arthritis Pain at Month 9 and 12
Description: as for outcome 20
Time Frame: Month 9, 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo Then CP-690,550 5 mg | Placebo Then CP-690,550 10 mg
Number analyzed (Participants) | 266 | 264 | 72 | 70
mm
  Month 9 | 32.06 (22.49) | 28.01 (20.81) | 28.97 (20.07) | 28.56 (22.74)
  Month 12 | 30.64 (22.03) | 27.94 (20.39) | 28.71 (23.05) | 28.20 (24.29)

22. Secondary Outcome: Physician Global Assessment (PGA) of Arthritis Pain at Baseline, Week 2, Month 1, 2, 3, 4.5 and 6
Description: Physician Global Assessment of Arthritis was measured on a 0 to 100 mm VAS, where 0 mm = very good and 100 mm = very bad.
Time Frame: Baseline, Week 2, Month 1, 2, 3, 4.5, 6
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 310 | 313 | 158
mm
  Baseline (n=310,313,158) | 60.48 (17.83) | 59.66 (17.03) | 58.87 (16.52)
  Week 2 (n=308,304,155) | 46.41 (20.14) | 43.79 (18.17) | 49.08 (18.90)
  Month 1 (n=302,303,154) | 38.35 (19.92) | 34.31 (18.70) | 42.86 (20.13)
  Month 2 (n=299,299,150) | 32.54 (19.36) | 29.40 (17.36) | 41.25 (20.42)
  Month 3 (n=293,292,148) | 31.97 (20.25) | 29.21 (19.31) | 39.54 (21.09)
  Month 4.5 (n=283,288,71) | 29.45 (19.84) | 26.11 (17.54) | 33.04 (21.06)
  Month 6 (n=278,280,68) | 25.83 (17.29) | 23.69 (16.62) | 27.88 (19.10)

23. Secondary Outcome: Physician Global Assessment (PGA) of Arthritis at Month 9 and 12
Description: as for outcome 22
Time Frame: Month 9, 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo Then CP-690,550 5 mg | Placebo Then CP-690,550 10 mg
Number analyzed (Participants) | 265 | 264 | 72 | 70
mm
  Month 9 | 24.36 (17.67) | 20.09 (14.23) | 22.70 (15.42) | 20.63 (17.35)
  Month 12 | 21.52 (17.14) | 18.12 (14.50) | 19.01 (15.01) | 17.59 (15.21)

24. Secondary Outcome: 36-Item Short-Form Health Survey (SF-36) at Baseline, Month 1, 3 and 6
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning) and is reported as 2 summary scores; physical component score and mental component score. Total score range for the summary scores = 0-100, where higher score represents higher level of functioning.
Time Frame: Baseline, Month 1, 3, 6
Population: FAS population included participants who received at least 1 dose of study medication. Here, 'n' is signifying those participants who were evaluable for the measure at given time points for each group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 312 | 315 | 158
units on a scale
  Baseline:physical functioning(n=312,315,158) | 32.53 (9.58) | 31.74 (9.62) | 32.76 (9.59)
  Baseline:role physical(n=312,315,158) | 33.73 (9.74) | 33.15 (9.43) | 33.91 (9.57)
  Baseline:social functioning(n=312,315,158) | 36.22 (11.15) | 37.04 (10.27) | 36.87 (11.63)
  Baseline:bodily pain(n=312,315,158) | 33.38 (7.25) | 33.94 (7.28) | 34.22 (7.47)
  Baseline:mental health(n=312,315,158) | 39.94 (12.52) | 41.05 (10.54) | 41.50 (11.38)
  Baseline:role emotional(n=312,315,158) | 35.51 (13.65) | 34.91 (13.00) | 35.36 (12.97)
  Baseline:vitality(n=312,315,158) | 40.84 (10.29) | 40.87 (8.89) | 41.33 (9.37)
  Baseline:general health(n=312,315,158) | 33.95 (9.14) | 34.27 (8.58) | 34.65 (8.32)
  Baseline:mental component(n=312,315,158) | 40.86 (12.59) | 41.56 (11.14) | 41.67 (11.57)
  Baseline:physical component(n=312,315,158) | 32.44 (7.82) | 32.02 (7.46) | 32.74 (7.60)
  Month 1:physical functioning(n=303,302,154) | 36.17 (10.33) | 36.71 (10.08) | 33.95 (9.72)
  Month 1:role physical(n=303,301,154) | 38.20 (10.33) | 39.00 (9.60) | 37.15 (9.41)
  Month 1:social functioning(n=303,302,154) | 40.25 (10.99) | 41.96 (9.73) | 39.29 (9.92)
  Month 1:bodily pain(n=303,302,154) | 39.02 (7.86) | 40.70 (7.69) | 36.87 (7.14)
  Month 1:mental health(n=303,302,153) | 43.40 (11.43) | 44.70 (10.00) | 42.79 (11.04)
  Month 1:role emotional(n=303,301,154) | 38.36 (12.79) | 39.27 (11.91) | 38.18 (12.97)
  Month 1:vitality(n=303,302,153) | 45.87 (10.17) | 46.71 (8.76) | 43.74 (9.00)
  Month 1:general health(n=303,302,154) | 37.86 (9.45) | 38.81 (8.65) | 36.39 (8.35)
  Month 1:mental component(n=303,301,153) | 44.04 (11.64) | 45.32 (10.13) | 43.80 (11.22)
  Month 1:physical component(n=303,301,153) | 37.12 (8.31) | 37.94 (7.96) | 34.86 (7.48)
  Month 3:physical functioning(n=294,291,147) | 37.15 (10.47) | 38.29 (10.60) | 34.35 (10.42)
  Month 3:role physical(n=294,292,147) | 39.25 (9.91) | 40.57 (9.69) | 36.50 (9.76)
  Month 3:social functioning(n=294,292,147) | 41.51 (10.46) | 42.44 (9.92) | 38.62 (11.04)
  Month 3:bodily pain(n=294,292,147) | 40.22 (8.24) | 41.82 (8.70) | 37.50 (8.26)
  Month 3:mental health(n=294,292,147) | 44.69 (10.45) | 45.15 (10.28) | 42.68 (10.88)
  Month 3:role emotional(n=293,291,146) | 38.36 (11.98) | 39.81 (12.04) | 37.42 (13.23)
  Month 3:vitality(n=294,292,147) | 47.05 (9.71) | 47.22 (9.05) | 43.84 (9.68)
  Month 3:general health(n=294,291,147) | 38.98 (9.69) | 39.45 (9.19) | 35.56 (9.37)
  Month 3:mental component(n=293,290,146) | 44.96 (10.75) | 45.35 (10.26) | 43.10 (11.12)
  Month 3:physical component(n=293,290,146) | 38.26 (8.46) | 39.53 (8.58) | 34.90 (8.37)
  Month 6:physical functioning(n=279,280,68) | 38.55 (10.60) | 39.42 (10.38) | 38.18 (9.63)
  Month 6:role physical(n=279,279,68) | 39.86 (9.82) | 41.02 (9.41) | 40.27 (8.86)
  Month 6:social functioning(n=279,280,68) | 41.97 (10.22) | 43.36 (10.01) | 43.67 (9.96)
  Month 6:bodily pain(n=279,280,68) | 41.01 (8.17) | 42.12 (8.45) | 41.91 (7.74)
  Month 6:mental health(n=279,280,68) | 44.43 (10.26) | 45.01 (10.27) | 44.12 (10.13)
  Month 6:role emotional(n=279,279,68) | 39.37 (12.11) | 40.49 (11.79) | 39.81 (12.38)
  Month 6:vitality(n=279,280,68) | 47.02 (9.82) | 47.80 (9.55) | 46.67 (8.93)
  Month 6:general health(n=279,280,68) | 40.03 (9.51) | 39.71 (9.17) | 38.10 (9.05)
  Month 6:mental component(n=279,279,68) | 44.73 (10.59) | 45.63 (10.29) | 45.13 (11.02)
  Month 6:physical component(n=279,279,68) | 39.49 (8.64) | 40.24 (8.43) | 39.24 (7.19)

25. Secondary Outcome: 36-Item Short-Form Health Survey (SF-36) at Month 9 and 12
Description: as for outcome 24
Time Frame: Month 9, 12
Population: FAS population included participants who received at least 1 dose of study medication. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n' signifies those participants who were evaluable for the measure at given time points for each group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo Then CP-690,550 5 mg | Placebo Then CP-690,550 10 mg
Number analyzed (Participants) | 267 | 264 | 72 | 70
units on a scale
  Month 9:physical functioning(n=267,263,72,70) | 39.40 (10.60) | 40.67 (10.12) | 38.86 (10.47) | 40.83 (9.76)
  Month 9:role physical(n=267,263,72,70) | 40.21 (9.99) | 42.03 (9.05) | 41.44 (9.70) | 42.99 (9.18)
  Month 9:social functioning(n=267,264,72,70) | 42.43 (9.97) | 43.67 (9.60) | 43.26 (11.23) | 44.11 (10.32)
  Month 9:bodily pain(n=267,264,72,70) | 41.83 (8.89) | 43.37 (8.45) | 42.31 (8.42) | 44.03 (8.26)
  Month 9:mental health(n=267,264,72,70) | 45.49 (10.69) | 46.03 (10.67) | 46.12 (10.49) | 45.11 (10.51)
  Month 9:role emotional(n=267,264,72,70) | 40.55 (11.54) | 42.16 (11.43) | 40.75 (12.67) | 41.02 (11.46)
  Month 9:vitality(n=267,264,72,70) | 48.39 (9.53) | 48.70 (9.41) | 48.38 (8.71) | 47.29 (10.43)
  Month 9:general health(n=266,264,72,70) | 39.77 (9.63) | 40.57 (9.29) | 40.38 (9.04) | 40.08 (9.50)
  Month 9:mental component(n=266,262,72,70) | 45.97 (10.45) | 46.61 (10.74) | 46.42 (11.01) | 45.22 (11.40)
  Month 9:physical component(n=266,262,72,70) | 39.79 (8.60) | 41.15 (8.15) | 40.07 (7.97) | 42.05 (6.93)
  Month 12:physical functioning(n=258, 250,70,67) | 39.07 (11.18) | 40.38 (10.24) | 38.61 (11.38) | 39.85 (10.97)
  Month 12:role physical(n=258, 250,70,67) | 40.51 (9.99) | 42.11 (9.31) | 42.51 (9.72) | 43.16 (9.51)
  Month 12:social functioning(n=258, 250,70,67) | 42.69 (10.14) | 43.63 (9.71) | 44.27 (9.72) | 44.36 (10.30)
  Month 12:bodily pain(n=258, 250,70,67) | 41.95 (8.77) | 43.28 (8.70) | 42.59 (9.07) | 45.49 (8.11)
  Month 12:mental health(n=258, 250,70,67) | 44.86 (10.63) | 45.52 (10.27) | 46.10 (10.81) | 45.65 (11.29)
  Month 12:role emotional(n=258, 250,70,67) | 40.02 (12.10) | 41.37 (11.79) | 42.92 (11.80) | 42.40 (11.92)
  Month 12:vitality(n=258, 250,70,67) | 48.08 (9.83) | 48.12 (9.22) | 49.77 (9.52) | 47.75 (10.45)
  Month 12:general health(n=258, 250,70,67) | 39.63 (9.64) | 39.88 (8.88) | 40.86 (9.34) | 39.43 (10.35)
  Month 12:mental component(n=258, 250,70,67) | 45.39 (10.69) | 45.92 (10.65) | 47.84 (11.04) | 46.33 (11.21)
  Month 12:physical component(n=258, 250,70,67) | 39.94 (8.83) | 41.13 (8.13) | 40.16 (9.14) | 41.62 (8.16)

26. Secondary Outcome: Medical Outcomes Study Sleep Scale (MOS-SS) at Baseline, Month 1, 3 and 6
Description: Participant-rated 12 item questionnaire to assess constructs of sleep over past week.7 subscales: sleep disturbance, snoring, awakened short of breath, sleep adequacy, somnolence (range:0-100); sleep quantity(range:0-24), optimal sleep(yes or no). 9 item index measures of sleep disturbance provide composite scores: sleep problem summary, overall sleep problem. Except Adequacy, Optimal, Quantity of sleep, higher scores=more impairment. Scores transformed(actual raw score(RS) minus lowest possible score divided by possible RS range*100);total score range:0-100,higher score=more intensity of attribute.
Time Frame: Baseline, Month 1, 3, 6
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 312 | 314 | 158
units on a scale
  Baseline:overall sleep problem(n=312,313,158) | 41.05 (20.68) | 40.89 (18.47) | 39.75 (18.25)
  Baseline:sleep problem summary(n=312,314,158) | 39.51 (21.22) | 40.08 (19.02) | 37.87 (18.37)
  Baseline:somnolence(n=312,314,158) | 34.38 (21.95) | 36.09 (21.59) | 34.94 (17.94)
  Baseline:snoring(n=310,314,157) | 32.26 (30.31) | 31.27 (31.27) | 33.76 (32.09)
  Baseline:quantity(n=312,313,158) | 6.88 (2.13) | 6.72 (1.55) | 6.82 (1.51)
  Baseline:sleep disturbance(n=312,313,158) | 44.39 (26.68) | 41.58 (24.61) | 41.20 (25.42)
  Baseline:awaken short of breath(n=312,314,158) | 18.91 (24.38) | 19.81 (24.38) | 17.34 (21.78)
  Baseline:adequacy(n=312,314,158) | 47.56 (28.78) | 44.97 (26.89) | 46.84 (25.69)
  Month 1:overall sleep problem(n=301,301,154) | 36.51 (19.94) | 34.77 (17.79) | 37.09 (18.02)
  Month 1:sleep problem summary(n=301,301,154) | 35.87 (20.50) | 34.45 (17.94) | 35.95 (18.32)
  Month 1:somnolence(n=301,302,154) | 31.58 (21.01) | 30.49 (20.05) | 33.33 (19.02)
  Month 1:snoring(n=300,302,153) | 29.87 (29.33) | 28.74 (30.29) | 32.03 (29.68)
  Month 1:quantity(n=301,301,154) | 6.90 (1.54) | 7.02 (1.55) | 6.81 (1.54)
  Month 1:sleep disturbance(n=301,302,154) | 38.43 (26.01) | 34.64 (24.20) | 37.42 (24.86)
  Month 1:awaken short of breath(n=301,301,154) | 18.34 (23.41) | 17.21 (21.91) | 14.94 (20.01)
  Month 1:adequacy(n=301,302,154) | 52.92 (27.91) | 51.52 (26.23) | 49.16 (23.51)
  Month 3:overall sleep problem(n=292,292,146) | 35.10 (18.58) | 34.06 (17.33) | 38.66 (17.32)
  Month 3:sleep problem summary(n=292,292,146) | 34.41 (19.04) | 33.80 (17.65) | 37.97 (17.21)
  Month 3:somnolence(n=292,292,146) | 30.07 (19.89) | 28.90 (18.75) | 35.43 (20.29)
  Month 3:snoring(n=290,292,144) | 31.31 (29.56) | 31.78 (30.23) | 31.81 (29.77)
  Month 3:quantity(n=293,292,147) | 6.87 (1.54) | 6.96 (1.46) | 6.76 (1.55)
  Month 3:sleep disturbance(n=292,292,146) | 36.67 (23.98) | 33.69 (23.01) | 37.77 (24.18)
  Month 3:awaken short of breath(n=292,292,146) | 19.38 (24.67) | 17.26 (21.19) | 18.08 (21.57)
  Month 3:adequacy(n=292,292,146) | 54.66 (27.42) | 51.58 (26.71) | 45.82 (25.54)
  Month 6:overall sleep problem(n=277,280,68) | 33.92 (19.36) | 33.11 (16.94) | 34.87 (18.29)
  Month 6:sleep problem summary(n=277,280,68) | 33.26 (19.87) | 33.30 (17.17) | 34.85 (18.81)
  Month 6:somnolence(n=277,280,68) | 31.12 (20.03) | 29.81 (18.23) | 30.29 (19.19)
  Month 6:snoring(n=271,280,68) | 31.14 (28.98) | 32.07 (29.21) | 31.47 (29.79)
  Month 6:quantity(n=278,279,68) | 6.86 (1.52) | 6.94 (1.42) | 6.82 (1.41)
  Month 6:sleep disturbance(n=277,280,68) | 34.48 (24.11) | 31.33 (21.96) | 34.78 (24.36)
  Month 6:awaken short of breath(n=277,280,68) | 17.62 (19.89) | 17.57 (20.87) | 17.06 (24.98)
  Month 6:adequacy(n=277,280,68) | 54.40 (28.34) | 51.64 (26.36) | 50.29 (26.76)

27. Secondary Outcome: Number of Participants With Optimal Sleep Assessed Using Medical Outcomes Study Sleep Scale (MOS-SS) at Baseline, Month 1, 3 and 6
Description: MOS-SS: participant-rated 12 item questionnaire to assess constructs of sleep over past week. It included 7 subscales: sleep disturbance, snoring, awakened short of breath, sleep adequacy, somnolence, sleep quantity and optimal sleep. Participants responded whether their sleep was optimal or not by choosing yes or no. Number of participants with optimal sleep are reported.
Time Frame: Baseline, Month 1, 3, 6
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 312 | 315 | 158
participants
  Baseline (n=312,315,158) | 139 | 139 | 70
  Month 1 (n=305,303,155) | 155 | 145 | 72
  Month 3 (n=294,292,147) | 139 | 152 | 65
  Month 6 (n=278,280,145) | 142 | 143 | 66

28. Secondary Outcome: Medical Outcome Study (MOS) Sleep Scale at Month 12
Description: as for outcome 26
Time Frame: Month 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo Then CP-690,550 5 mg | Placebo Then CP-690,550 10 mg
Number analyzed (Participants) | 258 | 249 | 70 | 66
units on a scale
  Overall sleep problem | 34.17 (18.71) | 32.24 (17.13) | 31.74 (17.41) | 33.58 (17.44)
  Sleep problem summary | 33.71 (19.11) | 32.58 (17.42) | 30.95 (17.09) | 32.53 (17.89)
  Somnolence | 29.30 (19.09) | 27.93 (17.70) | 30.86 (21.18) | 28.48 (15.45)
  Snoring | 30.32 (28.59) | 32.37 (29.70) | 31.43 (31.13) | 31.38 (27.58)
  Quantity | 6.94 (1.51) | 7.04 (1.30) | 6.83 (1.36) | 6.95 (1.42)
  Sleep disturbance | 34.78 (24.31) | 31.75 (21.95) | 29.41 (24.04) | 35.63 (22.81)
  Awaken short of breath | 19.77 (24.38) | 17.19 (21.25) | 17.71 (19.42) | 14.85 (17.30)
  Adequacy | 54.38 (26.14) | 53.29 (25.26) | 55.00 (25.01) | 55.76 (26.37)

29. Secondary Outcome: Number of Participants With Optimal Sleep Assessed Using Medical Outcomes Study Sleep Scale (MOS-SS) at Month 12
Description: as for outcome 27
Time Frame: Month 12
Population: as for outcome 11
Measure: Number; unit: participants
Groups:
- Placebo Then CP-690,550 5 mg: Placebo matched to CP-690,550 tablet orally twice daily for 3 to 6 months. Response was assessed at Month 3 and participants who failed to achieve at least 20% reduction in both swollen and tender joint counts from baseline, received CP-690,550 5 mg tablet orally twice daily up to Month 12. At Month 6, remaining participants received CP-690,550 5 mg tablet orally twice daily up to Month 12.
- Placebo Then CP-690,550 10 mg: Placebo matched to CP-690,550 tablet orally twice daily for 3 to 6 months. Response was assessed at Month 3 and participants who failed to achieve at least 20% reduction in both swollen and tender joint counts from baseline, received CP-690,550 10 mg tablet orally twice daily up to Month 12. At Month 6, remaining participants received CP-690,550 10 mg tablet orally twice daily up to Month 12.
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo Then CP-690,550 5 mg | Placebo Then CP-690,550 10 mg
Number analyzed (Participants) | 258 | 250 | 70 | 67
participants | 134 | 144 | 37 | 36

30. Secondary Outcome: Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale at Baseline, Month 1, 3, and 6
Description: FACIT-Fatigue is a 13-item questionnaire. Participant scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the participant's response to the questions (with the exception of 2 negatively stated), the greater the fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as 4 minus the participant's response. The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score). A higher score reflected an improvement in the participant's health status.
Time Frame: Baseline, Month 1, 3, 6
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 312 | 314 | 158
units on a scale
  Baseline (n=312,314,158) | 29.01 (11.01) | 28.65 (9.49) | 29.72 (8.97)
  Month 1 (n=301,302,153) | 33.16 (10.75) | 33.94 (8.91) | 31.78 (9.58)
  Month 3 (n=294,292,147) | 34.38 (10.07) | 34.99 (9.20) | 31.41 (9.95)
  Month 6 (n=277,280,68) | 35.14 (9.91) | 35.01 (9.45) | 35.24 (9.30)

31. Secondary Outcome: Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale at Month 12
Description: as for outcome 30
Time Frame: Month 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo Then CP-690,550 5 mg | Placebo Then CP-690,550 10 mg
Number analyzed (Participants) | 258 | 249 | 70 | 67
units on a scale | 35.02 (9.83) | 36.34 (9.15) | 36.93 (9.19) | 36.07 (9.64)

32. Secondary Outcome: Euro Quality of Life (EQ-5D)- Health State Profile Utility Score at Baseline, Month 3 and 6
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Baseline, Month 3, 6
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 311 | 314 | 158
units on a scale
  Baseline (n=311,314,158) | 0.46 (0.31) | 0.48 (0.29) | 0.51 (0.27)
  Month 3 (n=294,291,147) | 0.63 (0.24) | 0.68 (0.24) | 0.56 (0.28)
  Month 6 (n=277,280,68) | 0.66 (0.23) | 0.70 (0.21) | 0.65 (0.20)

33. Secondary Outcome: Euro Quality of Life (EQ-5D)- Health State Profile Utility Score at Month 12
Description: as for outcome 32
Time Frame: Month 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo Then CP-690,550 5 mg | Placebo Then CP-690,550 10 mg
Number analyzed (Participants) | 258 | 249 | 70 | 67
units on a scale | 0.68 (0.23) | 0.70 (0.21) | 0.66 (0.24) | 0.69 (0.23)

34. Other Pre Specified Outcome: Time to First Greater Than 1 Day Sequential Decrease in Pain From Baseline for Patient Global Assessment of Arthritis
Description: Patient global assessment of arthritis: participants answered: "Considering all the ways your arthritis affects you, how are you feeling today?" Participants responded by using a 0 - 100 mm VAS where 0 = very well and 100 = very poorly.
Time Frame: 2 weeks
Population: as for outcome 13
Measure: Number; unit: days
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 51 | 54 | 33
days | 3 | 3 | 3

35. Other Pre Specified Outcome: Time to First Greater Than 1 Day Sequential Decrease in Pain From Baseline for Patient Assessment of Arthritis Pain
Description: as for outcome 19
Time Frame: 2 weeks
Population: as for outcome 13
Measure: Number; unit: days
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 51 | 54 | 33
days | 3 | 3 | 3

36. Secondary Outcome: Work Limitations Questionnaire (WLQ) Score at Baseline, Month 3 and 6
Description: WLQ: participant-reported 25-item scale to evaluate degree to which health problems interfere with an ability to perform job roles along 4 dimensions: time management scale (5-items); physical demands scale (6-item); mental-interpersonal demands Scale (9-items); output demands scale (5-items). All the scales ranged from 0 (limited none of the time) to 100 (limited all of the time). Work loss index, which represented percentage of lost work over time period relative to a normative population, was derived (total score:0[no loss] to 100[complete loss of work]).
Time Frame: Baseline, Month 3, 6
Population: FAS population included participants who received at least 1 dose of study medication. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n' signifies those participants who were evaluable for each parameter at given time points for each group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 164 | 163 | 90
units on a scale
  Baseline:time management(n=152,149,80) | 47.13 (27.40) | 46.05 (27.83) | 39.98 (24.44)
  Baseline:physical demands(n=154,154,86) | 48.08 (25.92) | 50.83 (25.34) | 51.88 (24.98)
  Baseline:mental demands(n=158,154,83) | 36.58 (26.35) | 35.86 (25.72) | 30.31 (24.19)
  Baseline:output demands(n=153,149,79) | 41.93 (27.66) | 38.76 (28.34) | 32.72 (25.35)
  Baseline:work loss index(n=164,163,90) | 11.25 (6.04) | 10.76 (6.16) | 9.22 (5.28)
  Month 3:time management(n=139,131,69) | 38.56 (30.11) | 37.39 (30.53) | 36.99 (28.24)
  Month 3:physical demands(n=135, 32,66) | 43.14 (26.03) | 45.07 (30.63) | 52.78 (24.73)
  Month 3:mental demands(n=142,136,72) | 30.43 (27.99) | 31.60 (29.49) | 28.15 (23.69)
  Month 3:output demands(n=136,132,68) | 32.23 (27.77) | 33.43 (30.58) | 27.33 (24.32)
  Month 3:work loss index(n=145,138,73) | 9.29 (6.32) | 9.64 (7.10) | 8.77 (5.47)
  Month 6:time management(n=112,108,27) | 34.43 (28.40) | 35.73 (31.85) | 33.77 (31.88)
  Month 6:physical demands(n=114,110,24) | 48.72 (29.30) | 41.75 (30.91) | 48.13 (32.45)
  Month 6:mental demands(n=115,112,27) | 25.94 (26.35) | 27.98 (28.18) | 22.34 (26.57)
  Month 6:output demands(n=111,111,26) | 28.92 (26.55) | 28.98 (28.12) | 29.52 (29.09)
  Month 6:work loss index(n=116,114,28) | 8.73 (6.26) | 8.71 (6.64) | 8.03 (6.64)

37. Secondary Outcome: Work Limitations Questionnaire (WLQ) Score at Month 12
Description: as for outcome 36
Time Frame: Month 12
Population: FAS population included participants who received at least 1 dose of study medication. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n' signifies those participants who were evaluable for given parameters for each group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo Then CP-690,550 5 mg | Placebo Then CP-690,550 10 mg
Number analyzed (Participants) | 108 | 101 | 38 | 32
units on a scale
  Time management(n=105,98,35,31) | 37.01 (30.03) | 35.29 (31.80) | 30.82 (29.59) | 36.57 (30.80)
  Physical demands(n=105,97,36,28) | 44.15 (27.91) | 42.41 (31.59) | 47.15 (30.40) | 40.82 (30.86)
  Mental demands(n=108,100,36,32) | 27.27 (26.33) | 27.42 (27.56) | 20.70 (26.37) | 33.05 (29.78)
  Output demands(n=105,95,35,29) | 26.75 (25.54) | 25.67 (27.25) | 22.54 (25.05) | 28.43 (27.66)
  Work loss index(n=108,101,38,32) | 8.65 (6.12) | 8.28 (6.59) | 7.06 (5.81) | 8.89 (6.29)

38. Secondary Outcome: Work Productivity and Healthcare Resource Utilization (HCRU) at Baseline, Month 3 and 6
Description: Rheumatoid Arthritis (RA)-HCRU assessed healthcare usage during last 3 months for direct, indirect medical cost domains. Direct cost:visit to doctor, non-medical practitioner, nursing home, hospital, surgery, emergency room(ER) treatment, diagnostic tests, over-night stay, home healthcare services, aids/devices used. Indirect costs associated with functional disability:employment status, willingness to work, work disability due to RA, sick leave,part time work, ability to perform chores, chores done by family/friends/housekeeper. Assessment was based on 0 to 2-point scale;higher score=higher medical cost.
Time Frame: Baseline, Month 3, 6
Population: FAS population included participants who received at least 1 dose of study medication. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.'n' signifies those participants who were evaluable for each parameter at given time points for each group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 307 | 313 | 154
units on a scale
  Baseline:Seen any doctor(n=307,312,153) | 1.13 (0.34) | 1.11 (0.32) | 1.16 (0.37)
  Baseline:Treated in emergency room(n=307,313,154) | 1.94 (0.24) | 1.94 (0.23) | 1.95 (0.22)
  Baseline:Admitted for overnight stay(n=19,18,8) | 0.16 (0.37) | 0.22 (0.43) | 0.50 (0.93)
  Baseline:Hospitalization(n=307,313,154) | 1.95 (0.22) | 1.93 (0.26) | 1.94 (0.24)
  Baseline:Outpatient surgery(n=307,312,154) | 1.97 (0.16) | 1.98 (0.14) | 1.94 (0.24)
  Baseline:Non-study diagnostic test(n=307,312,154) | 1.85 (0.35) | 1.87 (0.33) | 1.86 (0.35)
  Baseline:In nursing home(n=307,312,154) | 2.00 (0.06) | 1.99 (0.08) | 1.99 (0.11)
  Baseline:Home healthcare services(n=307,312,154) | 1.99 (0.10) | 1.99 (0.11) | 1.99 (0.11)
  Baseline:Required aids/devices(n=307,311,154) | 1.88 (0.33) | 1.87 (0.34) | 1.88 (0.33)
  Baseline:Non-medical practitioner(n=307,312,154) | 1.96 (0.20) | 1.98 (0.14) | 1.98 (0.14)
  Baseline:Currently employed(n=307,312,154) | 1.64 (0.48) | 1.66 (0.47) | 1.62 (0.49)
  Baseline:Feel well enough to work(n=121,122,57) | 1.88 (0.33) | 1.89 (0.32) | 1.79 (0.41)
  Baseline:Unable to work due to RA(n=122,129,55) | 1.34 (0.48) | 1.25 (0.43) | 1.42 (0.50)
  Baseline:Lost job/retired early(n=121,116,54) | 1.64 (0.48) | 1.47 (0.50) | 1.50 (0.50)
  Baseline:Work disabled due to RA(n=126,120,53) | 1.50 (0.50) | 1.34 (0.48) | 1.47 (0.50)
  Baseline:Retired(n=132,133,59) | 1.50 (0.50) | 1.41 (0.49) | 1.41 (0.50)
  Baseline:Sick leave due to RA(n=286,278,145) | 1.75 (0.43) | 1.78 (0.41) | 1.81 (0.39)
  Baseline:Performed part time work(n=285,278,143) | 1.89 (0.31) | 1.89 (0.31) | 1.92 (0.28)
  Baseline:Performed paid work(n=287,277,144) | 1.67 (0.47) | 1.66 (0.47) | 1.66 (0.48)
  Baseline:Unable to do chores(n=305,307,153) | 1.44 (0.50) | 1.48 (0.50) | 1.44 (0.50)
  Baseline:Chores by housekeeper(n=306,312,154) | 1.85 (0.36) | 1.88 (0.32) | 1.88 (0.32)
  Baseline:Chores by family/friends(n=306,312,154) | 1.49 (0.50) | 1.49 (0.50) | 1.48 (0.50)
  Month 3:Seen any doctor(n=290,291,146) | 1.38 (0.49) | 1.41 (0.49) | 1.36 (0.48)
  Month 3:Treated in emergency room(n=290,291,146) | 1.96 (0.20) | 1.98 (0.15) | 1.96 (0.20)
  Month 3:Admitted for overnight stay(n=12,7,6) | 0.25 (0.62) | 0.14 (0.38) | 0.33 (0.82)
  Month 3:Hospitalization(n=288,291,146) | 1.99 (0.12) | 1.99 (0.12) | 1.97 (0.16)
  Month 3:Outpatient surgery(n=290,291,146) | 1.98 (0.14) | 1.98 (0.13) | 1.96 (0.20)
  Month 3:Non-study diagnostic test(n=288,291,146) | 1.91 (0.29) | 1.91 (0.29) | 1.90 (0.30)
  Month 3:In nursing home(n=290,291,146) | 2.00 (0.06) | 1.99 (0.08) | 2.00 (0.00)
  Month 3:Home healthcare services(n=289,291,146) | 1.99 (0.08) | 1.99 (0.12) | 1.99 (0.12)
  Month 3:Required aids/devices(n=288,291,146) | 1.91 (0.28) | 1.91 (0.29) | 1.81 (0.40)
  Month 3:Non-medical practitioner(n=290,291,146) | 1.98 (0.14) | 1.98 (0.14) | 1.99 (0.08)
  Month 3:Currently employed(n=289,291,146) | 1.64 (0.48) | 1.66 (0.48) | 1.63 (0.48)
  Month 3:Feel well enough to work(n=107,130,47) | 1.81 (0.39) | 1.75 (0.44) | 1.79 (0.41)
  Month 3:Unable to work due to RA(n=108,124,50) | 1.43 (0.50) | 1.49 (0.50) | 1.46 (0.50)
  Month 3:Lost job/retired early(n=109,125,49) | 1.58 (0.50) | 1.61 (0.49) | 1.55 (0.50)
  Month 3:Work disabled due to RA(n=108,123,47) | 1.49 (0.50) | 1.54 (0.50) | 1.51 (0.51)
  Month 3:Retired(n=132,129,57) | 1.45 (0.50) | 1.44 (0.50) | 1.39 (0.49)
  Month 3:Sick leave due to RA(n=265,266,139) | 1.88 (0.32) | 1.91 (0.28) | 1.83 (0.38)
  Month 3:Performed part time work(n=264,265,139) | 1.94 (0.24) | 1.96 (0.20) | 1.94 (0.23)
  Month 3:Performed paid work(n=265,266,139) | 1.72 (0.45) | 1.77 (0.42) | 1.72 (0.45)
  Month 3:Unable to do chores(n=284,286,147) | 1.65 (0.48) | 1.71 (0.46) | 1.57 (0.50)
  Month 3:Chores by housekeeper(n=289,290,146) | 1.90 (0.31) | 1.93 (0.25) | 1.93 (0.25)
  Month 3:Chores by family/friends(n=288,290,146) | 1.65 (0.48) | 1.68 (0.47) | 1.59 (0.49)
  Month 6:Seen any doctor(n=275,279,68) | 1.40 (0.49) | 1.37 (0.48) | 1.43 (0.50)
  Month 6:Treated in emergency room(n=275,279,68) | 1.95 (0.21) | 1.98 (0.15) | 1.97 (0.17)
  Month 6:Admitted for overnight stay (n=13,5,2) | 0.62 (0.87) | 0.40 (0.89) | 0.00 (0.00)
  Month 6:Hospitalization(n=274,279,68) | 1.97 (0.17) | 1.97 (0.16) | 2.00 (0.00)
  Month 6:Outpatient surgery(n=275,279,68) | 1.98 (0.13) | 1.98 (0.13) | 1.93 (0.26)
  Month 6:Non-study diagnostic test(n=274,279,68) | 1.91 (0.29) | 1.93 (0.25) | 1.85 (0.36)
  Month 6:In nursing home(n=275,279,68) | 2.00 (0.00) | 2.00 (0.00) | 2.00 (0.00)
  Month 6:Home healthcare services(n=273,278,68) | 1.99 (0.09) | 1.99 (0.08) | 2.00 (0.00)
  Month 6:Required aids/devices(n=274,278,68) | 1.91 (0.28) | 1.91 (0.29) | 1.93 (0.26)
  Month 6:Non-medical practitioner(n=275,279,68) | 1.99 (0.10) | 2.00 (0.06) | 2.00 (0.00)
  Month 6:Currently employed(n=274,279,68) | 1.65 (0.48) | 1.66 (0.47) | 1.65 (0.48)
  Month 6:Feel well enough to work(n=117,129,25) | 1.80 (0.40) | 1.71 (0.46) | 1.72 (0.46)
  Month 6:Unable to work due to RA(n=121,126,23) | 1.45 (0.50) | 1.49 (0.50) | 1.43 (0.51)
  Month 6:Lost job/retired early(n=118,125,23) | 1.63 (0.49) | 1.57 (0.50) | 1.52 (0.51)
  Month 6:Work disabled due to RA(n=117,125,23) | 1.53 (0.50) | 1.57 (0.50) | 1.65 (0.49)
  Month 6:Retired(n=129,136,30) | 1.47 (0.50) | 1.50 (0.50) | 1.47 (0.51)
  Month 6:Sick leave due to RA(n=250,255,59) | 1.92 (0.28) | 1.95 (0.23) | 1.93 (0.52)
  Month 6:Performed part time work(n=250,255,59) | 1.97 (0.17) | 1.97 (0.17) | 1.98 (0.13)
  Month 6:Performed paid work(n=249,255,59) | 1.78 (0.41) | 1.81 (0.39) | 1.76 (0.43)
  Month 6:Unable to do chores(n=269,276,67) | 1.70 (0.46) | 1.73 (0.45) | 1.69 (0.47)
  Month 6:Chores by housekeeper(n=275,277,68) | 1.90 (0.30) | 1.95 (0.22) | 1.91 (0.29)
  Month 6:Chores by family/friends(n=274,277,68) | 1.71 (0.46) | 1.75 (0.43) | 1.79 (0.41)

39. Secondary Outcome: Work Productivity and Healthcare Resource Utilization (HCRU) at Month 12
Description: Rheumatoid Arthritis (RA)-HCRU assessed healthcare usage during last 3 months for direct, indirect medical cost domains. Direct cost:visit to doctor,non-medical practitioner,nursing home,hospital,surgery,emergency room(ER) treatment,diagnostic tests, over-night stay,home healthcare services, aids/devices used. Indirect costs associated with functional disability:employment status,willingness to work,work disability due to RA,sick leave,part time work,ability to perform chores,chores done by family/friends/housekeeper. Assessment was based on 0 to 2-point scale;higher score=higher medical cost.
Time Frame: Month 12
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo Then CP-690,550 5 mg | Placebo Then CP-690,550 10 mg
Number analyzed (Participants) | 254 | 246 | 70 | 66
units on a scale
  Seen any doctor(n=254,243,70,66) | 1.48 (0.50) | 1.44 (0.50) | 1.40 (0.49) | 1.50 (0.50)
  Treated in ER(n=254,246,70,67) | 1.95 (0.22) | 1.95 (0.22) | 1.91 (0.28) | 1.93 (0.26)
  Admitted for overnight stay (n=13,12,6,5) | 0.23 (0.60) | 0.25 (0.62) | 0.33 (0.82) | 0.00 (0.00)
  Hospitalization(n=254,246,70,67) | 1.97 (0.17) | 1.97 (0.16) | 1.99 (0.16) | 1.97 (0.12)
  Had outpatient surgery(n=253,246,70,67) | 1.97 (0.18) | 1.98 (0.14) | 1.97 (0.17) | 1.97 (0.17)
  Diagnostic test(n=253,246,70,67) | 1.87 (0.33) | 1.90 (0.30) | 1.91 (0.28) | 1.84 (0.37)
  In nursing home(n=254,245,70,67) | 1.98 (0.12) | 2.00 (0.00) | 2.00 (0.00) | 2.00 (0.00)
  Home healthcare services(n=252,246,70,67) | 2.00 (0.06) | 2.00 (0.06) | 1.99 (0.12) | 2.00 (0.00)
  Required aids/devices(n=254,246,70,67) | 1.92 (0.28) | 1.93 (0.25) | 1.94 (0.23) | 1.93 (0.26)
  Non-medical practitioner(n=254,246,70,67) | 1.99 (0.09) | 1.99 (0.11) | 1.96 (0.20) | 2.00 (0.00)
  Currently employed(n=254,246,70,67) | 1.66 (0.47) | 1.65 (0.48) | 1.50 (0.50) | 1.63 (0.49)
  Feel well enough to work(n=102,107,18,19) | 1.74 (0.44) | 1.64 (0.48) | 1.72 (0.46) | 1.74 (0.45)
  Unable to work due to RA(n=100,107,19,19) | 1.50 (0.50) | 1.54 (0.50) | 1.37 (0.50) | 1.63 (0.50)
  Lost job/retired early(n=99,103,18,19) | 1.62 (0.49) | 1.55 (0.50) | 1.56 (0.51) | 1.58 (0.51)
  Work disabled due to RA(n=103,106,18,19) | 1.57 (0.50) | 1.56 (0.50) | 1.39 (0.50) | 1.58 (0.51)
  Retired(n=114,117,22,22) | 1.42 (0.50) | 1.44 (0.50) | 1.36 (0.49) | 1.32 (0.48)
  Sick leave due to RA(n=223,215,65,59) | 1.93 (0.25) | 1.94 (0.24) | 1.98 (0.12) | 1.93 (0.25)
  Performed part time work(n=224,217,64,57) | 1.96 (0.19) | 1.97 (0.18) | 1.98 (0.13) | 1.96 (0.19)
  Performed paid work(n=224,222,64,57) | 1.78 (0.41) | 1.76 (0.43) | 1.72 (0.45) | 1.75 (0.43)
  Unable to do chores(n=250,246,69,66) | 1.73 (0.44) | 1.77 (0.42) | 1.74 (0.44) | 1.89 (0.31)
  Chores by housekeeper(n=254,246,70,67) | 1.91 (0.29) | 1.96 (0.19) | 2.00 (0.00) | 1.93 (0.26)
  Chores by family/friends(n=253,246,70,66) | 1.75 (0.43) | 1.80 (0.40) | 1.79 (0.41) | 1.82 (0.39)

40. Secondary Outcome: Number of Events Including Visits, Surgeries, Tests or Devices as Assessed Using RA-HCRU at Baseline, Month 3 and 6
Description: RA-HCRU assessed healthcare usage during previous 3 months for direct or indirect medical cost domains. Any RA/non-RA related number of events including visits to doctor, non-medical practitioner, hospital ER treatment, hospitalizations, number of surgeries, diagnostic tests, and devices/aids used were reported.
Time Frame: Baseline, Month 3, 6
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: events
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 266 | 280 | 130
events
  Baseline:Doctor visit(n=266,280,130) | 4.27 (3.99) | 4.17 (3.58) | 4.13 (3.80)
  Baseline:RA related doctor visit(n=266,280,130) | 1.33 (0.85) | 1.32 (0.71) | 1.25 (0.61)
  Baseline:Hospital ER visit(n=19,18,8) | 1.26 (0.81) | 1.28 (0.67) | 1.38 (0.74)
  Baseline:RA related ER visit(n=19,18,8) | 0.58 (0.77) | 0.50 (0.51) | 0.88 (0.83)
  Baseline:Hospitalization(n=16,23,9) | 1.50 (2.00) | 1.26 (0.45) | 1.22 (0.67)
  Baseline:RA related hospitalization(n=16,23,9) | 0.94 (0.68) | 1.09 (0.90) | 0.78 (0.67)
  Baseline:Outpatient surgery(n=8,6,9) | 1.13 (0.35) | 1.17 (0.41) | 1.33 (0.50)
  Baseline:RA related outpatient surgery(n=8,5,9) | 0.88 (0.64) | 0.20 (0.45) | 0.56 (0.88)
  Baseline:Non-study diagnostic test(n=45,39,22) | 1.64 (1.03) | 2.13 (2.34) | 1.64 (0.95)
  Baseline:RA related diagnostic test(n=45,40,22) | 0.80 (0.87) | 0.90 (0.98) | 0.73 (0.88)
  Baseline:Non-medical practitioner visit(n=13,6,3) | 8.08 (7.90) | 2.83 (1.83) | 8.00 (2.00)
  Baseline:RA related non-medical visit(n=13,6,3) | 1.23 (0.73) | 1.00 (0.89) | 1.33 (0.58)
  Month 3:Doctor visit(n=183,174,94) | 4.50 (4.18) | 4.05 (3.77) | 4.66 (4.94)
  Month 3:RA related doctor visit(n=183,174,94) | 1.06 (0.75) | 0.97 (0.72) | 1.03 (0.71)
  Month 3:Hospital ER visit(n=11,7,6) | 1.36 (0.92) | 1.00 (0.00) | 1.17 (0.41)
  Month 3:RA related ER visit(n=12,7,6) | 0.17 (0.39) | 0.29 (0.76) | 0.00 (0.00)
  Month 3:Hospitalization(n=4,4,4) | 1.00 (0.00) | 1.00 (0.00) | 0.75 (0.50)
  Month 3:RA related hospitalization(n=4,4,4) | 0.25 (0.50) | 0.50 (0.58) | 0.25 (0.50)
  Month 3:Outpatient surgery(n=6,5,6) | 2.17 (1.94) | 1.00 (0.00) | 1.00 (0.00)
  Month 3:RA related outpatient surgery(n=6,5,6) | 0.00 (0.00) | 0.00 (0.00) | 0.17 (0.41)
  Month 3:Non-study diagnostic test(n=24,26,15) | 1.63 (1.21) | 1.35 (0.63) | 1.33 (0.82)
  Month 3:RA related diagnostic test(n=26,27,15) | 0.23 (0.65) | 0.22 (0.51) | 0.47 (0.52)
  Month 3:Non-medical practitioner visit(n=6,6,1) | 4.00 (2.28) | 3.00 (3.52) | 40.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.
  Month 3:RA related non-medical visit(n=6,6,1) | 0.67 (1.03) | 0.67 (0.52) | 4.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.
  Month 6:Doctor visit(n=168,178,39) | 3.54 (3.87) | 3.07 (2.73) | 3.08 (3.96)
  Month 6:RA related doctor visit(n=168,177,39) | 0.91 (0.65) | 0.97 (0.71) | 0.74 (0.59)
  Month 6:Hospital ER visit(n=13,4,2) | 1.31 (0.63) | 1.00 (0.00) | 2.50 (2.12)
  Month 6:RA related ER visit(n=13,6,2) | 0.08 (0.28) | 0.00 (0.00) | 0.00 (0.00)
  Month 6:Hospitalization(n=8,5,2) | 1.13 (0.35) | 1.00 (0.00) | 1.00 (0.00)
  Month 6:RA related hospitalization(n=8,7,2) | 0.38 (0.74) | 0.29 (0.76) | 1.00 (0.00)
  Month 6:Outpatient surgery(n=5,5,5) | 1.00 (0.00) | 1.40 (0.55) | 1.00 (0.00)
  Month 6:RA related outpatient surgery(n=5,5,5) | 0.00 (0.00) | 0.00 (0.00) | 0.20 (0.45)
  Month 6:Non-study diagnostic test(n=23,20,9) | 2.04 (1.49) | 1.60 (1.10) | 1.11 (0.33)
  Month 6:RA related diagnostic test(n=25,20,10) | 0.28 (0.54) | 0.35 (0.67) | 0.20 (0.42)
  Month 6:Non-medical practitioner visit(n=3,1,1) | 12.67 (11.02) | 12.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter
  Month 6:RA related non-medical visit(n=3,1,1) | 0.33 (0.58) | 4.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter

41. Secondary Outcome: Number of Events Including Visits, Surgeries, Tests or Devices as Assessed Using RA-HCRU at Month 12
Description: as for outcome 40
Time Frame: Month 12
Population: FAS population included participants who received at least 1 dose of study medication. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n' signifies those participants who were evaluable for this measure for given parameters for each group respectively.
Measure: Mean (Standard Deviation); unit: events
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo Then CP-690,550 5 mg | Placebo Then CP-690,550 10 mg
Number analyzed (Participants) | 136 | 139 | 42 | 34
events
  Doctor visit(n=136,139,42,34) | 3.17 (3.59) | 2.58 (2.62) | 3.19 (4.58) | 2.62 (1.65)
  RA related doctor visit (n=136,139,42,34) | 0.89 (0.66) | 0.74 (0.64) | 1.05 (0.82) | 0.79 (0.69)
  Hospital ER visit(n=13,12,6,5) | 1.15 (0.38) | 1.17 (0.58) | 1.67 (1.63) | 1.00 (0.00)
  RA related ER visit(n=13,12,6,5) | 0.15 (0.55) | 0.33 (0.65) | 0.33 (0.82) | 0.00 (0.00)
  Hospitalization(n=7,8,1,2) | 1.00 (0.00) | 1.00 (0.00) | 1.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | 1.50 (0.71)
  RA related hospitalization(n=8,8,1,2) | 0.50 (0.93) | 0.63 (0.92) | 0.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | 0.00 (0.00)
  Outpatient surgery(n=4,5,2,2) | 1.25 (0.50) | 1.60 (1.34) | 1.00 (0.00) | 1.00 (0.00)
  RA related outpatient surgery(n=8,5,2,2) | 0.13 (0.35) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Non-study diagnostic test(n=30,25,6,9) | 1.67 (0.88) | 1.68 (1.44) | 1.33 (0.52) | 2.00 (0.87)
  RA related diagnostic test(n=32,25,6,11) | 0.34 (0.70) | 0.12 (0.33) | 0.00 (0.00) | 0.09 (0.30)
  Non-medical practitioner visit(n=2,2,3,0) | 3.00 (1.41) | 6.00 (2.83) | 3.00 (2.65) | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter.
  RA related non-medical visit(n=2,3,3,0) | 0.00 (0.00) | 0.67 (0.58) | 0.67 (0.58) | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter.

42. Secondary Outcome: Number of Days as Assessed Using RA-HCRU at Baseline, Month 3 and 6
Description: RA-HCRU assessed healthcare usage during previous 3 months for direct or indirect medical cost domains.Any RA or non-RA related number of days spent in hospital, nursing home, aids/devices used, on sick leave, work per week, performed part time work, performed paid work, chores done by housekeeper and chores done by family/friends.
Time Frame: Baseline, Month 3, 6
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 154 | 158 | 78
days
  Baseline:Hospital length of stay(n=16,23,8) | 12.69 (6.05) | 15.26 (13.03) | 14.50 (15.97)
  Baseline:Days in nursing home(n=1,2,1) | 28.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | 14.50 (0.71) | 21.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.
  Baseline:Days aids/devices used(n=37,40,19) | 84.92 (71.64) | 100.78 (109.26) | 65.37 (74.55)
  Baseline:RA related aids used(n=37,42,19) | 1.65 (1.18) | 1.90 (1.36) | 1.42 (0.84)
  Baseline:Days of work per week(n=110,106,59) | 5.02 (1.05) | 5.01 (0.88) | 4.86 (1.02)
  Baseline:Days on sick leave due to RA(n=71,61,27) | 27.06 (33.38) | 30.26 (35.56) | 31.41 (32.27)
  Baseline:Days of part time work(n=30,29,12) | 22.77 (28.95) | 20.86 (29.44) | 34.83 (34.89)
  Baseline:Paid work, bothered by RA(n=94,93,48) | 40.11 (30.69) | 39.26 (29.85) | 43.15 (32.11)
  Baseline:Chores by housekeeper(n=46,37,18) | 27.17 (35.34) | 19.73 (28.01) | 37.28 (38.31)
  Baseline:Chores by family(n=154,158,79) | 41.26 (38.38) | 34.92 (33.94) | 37.81 (35.78)
  Month 3:Hospital length of stay(n=4,4,4) | 7.00 (4.24) | 8.25 (2.99) | 3.75 (0.50)
  Month 3:Days in nursing home(n=1,2,0) | 10.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | 14.00 (9.90) | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter.
  Month 3:Days aids/devices used(n=24,28,28) | 104.96 (87.40) | 104.36 (128.12) | 120.75 (152.78)
  Month 3:RA related aids used(n=25,28,28) | 1.68 (0.95) | 1.68 (1.39) | 1.79 (1.69)
  Month 3:Days of work per week(n=104,99,52) | 5.16 (1.01) | 5.12 (1.08) | 4.94 (1.00)
  Month 3:Days on sick leave due to RA(n=31,22,24) | 28.23 (34.67) | 28.45 (39.07) | 24.58 (33.18)
  Month 3:Days of part time work(n=16,11,8) | 20.06 (28.06) | 36.91 (37.77) | 36.13 (31.16)
  Month 3:Paid work, bothered by RA(n=75,62,38) | 31.25 (33.22) | 33.15 (30.42) | 42.32 (31.88)
  Month 3:Chores by housekeeper(n=30,19,10) | 26.87 (34.10) | 16.58 (26.03) | 21.40 (26.42)
  Month 3:Chores by family(n=97,92,60) | 34.23 (34.27) | 30.51 (33.93) | 41.92 (36.89)
  Month 6:Hospital length of stay(n=8,7,2) | 9.63 (7.76) | 6.43 (5.03) | 13.50 (0.71)
  Month 6:Days in nursing home(n=0,0,0) | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter. | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter. | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter.
  Month 6:Days aids/devices used(n=23,26,5) | 135.04 (104.11) | 116.27 (130.92) | 129.20 (42.11)
  Month 6:RA related aids used(n=24,26,5) | 1.79 (1.18) | 1.85 (1.43) | 1.80 (1.48)
  Month 6:Days of work per week(n=92,95,24) | 5.15 (1.04) | 5.04 (0.94) | 4.88 (0.99)
  Month 6:Days on sick leave due to RA(n=21,14,4) | 27.71 (36.77) | 24.43 (31.00) | 10.75 (13.45)
  Month 6:Days of part time work(n=7,8,2) | 35.43 (27.85) | 28.00 (36.01) | 7.50 (3.54)
  Month 6:Paid work, bothered by RA(n=54,46,13) | 30.80 (31.45) | 31.74 (30.04) | 33.31 (30.18)
  Month 6:Chores by housekeeper(n=26,13,6) | 22.42 (28.69) | 20.92 (31.17) | 43.50 (41.56)
  Month 6:Chores by family(n=78,68,14) | 29.53 (31.60) | 24.90 (31.36) | 33.93 (37.88)

43. Secondary Outcome: Number of Days as Assessed Using RA-HCRU at Month 12
Description: as for outcome 42
Time Frame: Month 12
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo Then CP-690,550 5 mg | Placebo Then CP-690,550 10 mg
Number analyzed (Participants) | 86 | 84 | 34 | 23
days
  Hospital length of stay(n=8,8,1,2) | 8.88 (6.73) | 12.38 (11.98) | 2.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | 1.50 (0.71)
  Days in nursing home(n=4,0,0,0) | 19.50 (8.35) | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter. | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter. | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter.
  Days aids/devices used(n=19,15,4,5) | 111.79 (84.57) | 161.40 (382.20) | 225.00 (155.88) | 62.00 (75.38)
  RA related aids used(n=21,16,4,5) | 1.19 (1.21) | 2.50 (4.76) | 2.50 (1.73) | 1.80 (1.30)
  Days of work per week(n=86,84,34,23) | 5.20 (1.03) | 5.35 (0.74) | 5.00 (1.10) | 5.22 (0.80)
  Days on sick leave due to RA(n=15,12,1,4) | 36.40 (42.27) | 13.58 (25.37) | 20.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | 31.00 (41.49)
  Days of part time work(n=8,7,1,2) | 14.88 (30.48) | 6.71 (3.15) | 24.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | 52.50 (53.03)
  Paid work, bothered by RA(n=49,53,18,14) | 39.08 (35.44) | 40.02 (33.50) | 40.39 (34.19) | 47.57 (39.16)
  Chores by housekeeper(n=23,9,0,5) | 32.17 (36.69) | 17.22 (28.01) | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter. | 6.60 (3.29)
  Chores by family(n=63,48,14,12) | 26.67 (32.49) | 24.98 (29.88) | 26.43 (32.22) | 26.00 (31.05)

44. Secondary Outcome: Number of Hours Per Day as Assessed RA-HCRU at Baseline, Month 3 and 6
Description: RA-HCRU assessed healthcare usage during previous 3 months for direct or indirect medical cost domains. Any RA or non-RA related number of hours spent per day for home healthcare services, chores done by housekeeper, chores done by family or friends, work done and work missed were reported.
Time Frame: Baseline, Month 3, 6
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 154 | 159 | 79
hours per day
  Baseline:Home healthcare services (n=3,4,2) | 4.67 (6.35) | 2.75 (2.36) | 1.50 (0.71)
  Baseline:RA related home HC services(n=3,4,2) | 0.67 (0.58) | 1.00 (0.82) | 0.50 (0.71)
  Baseline:Work done(n=110,106,59) | 7.84 (2.85) | 7.45 (2.27) | 7.24 (1.89)
  Baseline:Missed work due to RA(n=30,29,12) | 4.30 (4.18) | 6.24 (16.81) | 7.33 (8.07)
  Baseline:Chores by housekeeper(n=46,37,18) | 4.61 (3.96) | 4.62 (2.78) | 5.17 (5.15)
  Baseline:Chores by family(n=154,159,79) | 4.27 (4.81) | 3.86 (7.09) | 4.30 (5.59)
  Month 3:Home healthcare services(n=2,4,2) | 1.50 (0.71) | 3.25 (2.06) | 1.50 (0.71)
  Month 3:RA related home HC services(n=2,4,2) | 0.00 (0.00) | 0.25 (2.50) | 1.00 (1.41)
  Month 3:Work done(n=104,98,53) | 8.99 (7.48) | 7.64 (2.20) | 8.06 (4.94)
  Month 3:Missed work due to RA(n=16,11,8) | 3.94 (1.88) | 4.18 (2.14) | 3.88 (1.13)
  Month 3:Chores by housekeeper(n=30,19,10) | 4.17 (2.68) | 3.74 (3.74) | 3.30 (2.00)
  Month 3:Chores by family(n=98,89,59) | 3.32 (3.30) | 2.98 (3.35) | 4.97 (5.77)
  Month 6:Home healthcare services(n=2,2,0) | 17.00 (9.90) | 2.00 (1.41) | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter.
  Month 6:RA related home HC services(n=2,2,0) | 1.00 (1.41) | 2.00 (1.41) | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter.
  Month 6:Work done(n=92,95,24) | 8.12 (1.89) | 7.53 (1.72) | 8.50 (5.34)
  Month 6:Missed work due to RA(n=7,8,1) | 4.43 (1.62) | 3.38 (1.69) | 2.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.
  Month 6:Chores by housekeeper(n=25,13,6) | 4.64 (3.01) | 5.69 (6.45) | 5.17 (3.13)
  Month 6:Chores by family(n=77,66,14) | 3.73 (3.58) | 2.91 (3.30) | 4.36 (2.68)

45. Secondary Outcome: Number of Hours Per Day as Assessed RA-HCRU at Month 12
Description: as for outcome 44
Time Frame: Month 12
Population: FAS population included participants who received at least 1 dose of study medication. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.'n' signifies those participants who were evaluable for given parameters for each group respectively.
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo Then CP-690,550 5 mg | Placebo Then CP-690,550 10 mg
Number analyzed (Participants) | 85 | 85 | 34 | 24
hours per day
  Home healthcare services(n=1,1,1,0) | 1.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | 2.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | 1.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter.
  RA related healthcare services(n=1,1,1,0) | 0.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | 2.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | 1.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter.
  Work done(n=85,85,34,24) | 8.60 (4.00) | 7.67 (1.77) | 8.79 (5.85) | 7.38 (1.86)
  Missed work due to RA(n=8,7,1,2) | 5.00 (6.21) | 3.29 (1.80) | 0.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | 4.00 (1.41)
  Chores by housekeeper(n=22,9,0,5) | 4.86 (2.71) | 3.89 (1.96) | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter. | 4.40 (2.30)
  Chores by family(n=62,47,14,12) | 3.24 (3.26) | 2.70 (2.22) | 2.50 (1.40) | 5.92 (8.08)

46. Secondary Outcome: Work Performance in Past 3 Months on Days Bothered as Assessed Using RA-HCRU at Baseline, Month 3 and 6
Description: Work performance of participants on number of days bothered was based on a 0 to 10-point scale, where higher score indicated lower work performance.
Time Frame: Baseline, Month 3, 6
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 239 | 238 | 124
units on a scale
  Baseline (n=239, 238, 119) | 5.03 (5.89) | 4.72 (3.22) | 4.55 (3.14)
  Month 3 (n= 223, 229, 124) | 3.74 (3.04) | 3.18 (3.21) | 3.97 (3.15)
  Month 6 (n= 210, 224, 46) | 3.40 (3.06) | 2.66 (2.83) | 3.24 (2.86)

47. Secondary Outcome: Work Performance in Past 3 Months on Days Bothered as Assessed Using RA-HCRU at Month 12
Description: as for outcome 46
Time Frame: Month 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo Then CP-690,550 5 mg | Placebo Then CP-690,550 10 mg
Number analyzed (Participants) | 174 | 180 | 50 | 50
units on a scale | 2.79 (2.67) | 2.52 (2.74) | 2.84 (2.13) | 3.08 (2.60)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- CP-690,550 5 mg (Up To Month 3): CP-690,550 5 mg Film-coated tablet administered orally twice daily up to Month 3.
- CP-690,550 10 mg (Up To Month 3): CP-690,550 10 mg Film-coated tablet administered orally twice daily up to Month 3.
- Placebo (Up To Month 3): Matching placebo Film-coated tablet orally twice daily up to Month 3.
- CP-690,550 5 mg (Month 3 to 6): CP-690,550 5 mg twice daily from Month 3 to 6.
- CP-690,550 10 mg (Month 3 to 6): CP-690,550 10 mg tablet twice daily from Month 3 to 6.
- Placebo (Month 3 to 6): Matching placebo twice daily from Month 3 to 6.
- Placebo, Then CP-690,550 5 mg (Month 3 to 6): Participants who received matching placebo twice daily up to Month 3, received CP-690,550 5 mg tablet twice daily from Month 3 to 6.
- Placebo, Then CP-690,550 10 mg (Month 3 to 6): Participants who received matching placebo twice daily up to Month 3, received CP-690,550 10 mg tablet twice daily from Month 3 to 6.
- CP-690,550 5 mg (Post Month 6): CP-690,550 5 mg tablet orally twice daily from Month 6 to Month 12.
- CP-690,550 10 mg (Post Month 6): CP-690,550 10 mg tablet orally twice daily from Month 6 to 12.
- Placebo, Then CP-690,550 5 mg (Post Month 6): Participants who received matching placebo twice daily up to Month 3 and matching placebo or CP-690,550 5 mg tablet orally twice daily from Month 3 to 6, received CP-690,550 5 mg tablet twice daily from Month 6 to 12.
- Placebo, Then CP-690,550 10 mg (Post Month 6): Participants who received matching placebo twice daily up to Month 3 and matching placebo or CP-690,550 10 mg tablet orally twice daily from Month 3 to 6, received CP-690,550 10 mg tablet twice daily from Month 6 to 12.
Arm/Group | CP-690,550 5 mg (Up To Month 3) | CP-690,550 10 mg (Up To Month 3) | Placebo (Up To Month 3) | CP-690,550 5 mg (Month 3 to 6) | CP-690,550 10 mg (Month 3 to 6) | Placebo (Month 3 to 6) | Placebo, Then CP-690,550 5 mg (Month 3 to 6) | Placebo, Then CP-690,550 10 mg (Month 3 to 6) | CP-690,550 5 mg (Post Month 6) | CP-690,550 10 mg (Post Month 6) | Placebo, Then CP-690,550 5 mg (Post Month 6) | Placebo, Then CP-690,550 10 mg (Post Month 6)
Serious Adverse Events (participants affected / at risk) | 9/315 | 8/318 | 6/159 | 5/315 | 7/318 | 0/81 | 0/38 | 0/40 | 7/315 | 9/318 | 2/79 | 0/80
Other Adverse Events (participants affected / at risk) | 95/315 | 89/318 | 51/159 | 69/315 | 73/318 | 12/81 | 16/38 | 18/40 | 32/315 | 47/318 | 15/79 | 17/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 5 mg (Up To Month 3) (N=315) | CP-690,550 10 mg (Up To Month 3) (N=318) | Placebo (Up To Month 3) (N=159) | CP-690,550 5 mg (Month 3 to 6) (N=315) | CP-690,550 10 mg (Month 3 to 6) (N=318) | Placebo (Month 3 to 6) (N=81) | Placebo, Then CP-690,550 5 mg (Month 3 to 6) (N=38) | Placebo, Then CP-690,550 10 mg (Month 3 to 6) (N=40) | CP-690,550 5 mg (Post Month 6) (N=315) | CP-690,550 10 mg (Post Month 6) (N=318) | Placebo, Then CP-690,550 5 mg (Post Month 6) (N=79) | Placebo, Then CP-690,550 10 mg (Post Month 6) (N=80)
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic foot infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster disseminated (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiectasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Salivary gland calculus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia cryptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 5 mg (Up To Month 3) (N=315) | CP-690,550 10 mg (Up To Month 3) (N=318) | Placebo (Up To Month 3) (N=159) | CP-690,550 5 mg (Month 3 to 6) (N=315) | CP-690,550 10 mg (Month 3 to 6) (N=318) | Placebo (Month 3 to 6) (N=81) | Placebo, Then CP-690,550 5 mg (Month 3 to 6) (N=38) | Placebo, Then CP-690,550 10 mg (Month 3 to 6) (N=40) | CP-690,550 5 mg (Post Month 6) (N=315) | CP-690,550 10 mg (Post Month 6) (N=318) | Placebo, Then CP-690,550 5 mg (Post Month 6) (N=79) | Placebo, Then CP-690,550 10 mg (Post Month 6) (N=80)
Anaemia (Blood and lymphatic system disorders) | 7 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 14 | 10 | 6 | 0 | 0 | 0 | 0 | 0 | 6 | 1 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 4 | 8 | 2 | 4 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 8 | 6 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 11 | 8 | 4 | 6 | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 7 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 6 | 3 | 4 | 3 | 4 | 3 | 0 | 1 | 3 | 6 | 2 | 2
Nasopharyngitis (Infections and infestations) | 16 | 7 | 12 | 6 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 3 | 5 | 5 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 19 | 23 | 7 | 13 | 9 | 0 | 1 | 3 | 11 | 18 | 3 | 3
Alanine aminotransferase increased (Investigations) | 6 | 6 | 4 | 1 | 5 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 8 | 0 | 2 | 3 | 2 | 0 | 1 | 3 | 2 | 3 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 12 | 10 | 6 | 2 | 5 | 2 | 1 | 0 | 0 | 5 | 2 | 0
Hypertension (Vascular disorders) | 4 | 7 | 1 | 3 | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oesophageal spasm (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Device connection issue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 4 | 8 | 1 | 3 | 0 | 2 | 2 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0
Abscess jaw (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis infected (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 7 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 2 | 3 | 2 | 0 | 0 | 5 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 5 | 5 | 1 | 1 | 2 | 3 | 7 | 0 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 3 | 5 | 0 | 1 | 1 | 3 | 7 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 5 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 2 | 0 | 3 | 2 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 2 | 4 | 4 | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.